

Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Demonstrate Lot-to-Lot Consistency of 3 Lots of a Tetravalent Dengue Vaccine Candidate in Healthy Adults in Non-Endemic Country(ies) for Dengue

NCT Number: NCT03423173

Protocol Approve Date: 29 October 2018

Certain information within this protocol has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information (PPD) or company confidential information (CCI).

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.



### **PROTOCOL**

A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Demonstrate Lot-to-Lot Consistency of 3 Lots of a Tetravalent Dengue Vaccine Candidate in Healthy Adults in Non-Endemic Country(ies) for Dengue

# Lot-to-lot Consistency of 3 Lots of TDV in Non-Endemic Country(ies) for Dengue

**Sponsor:** Takeda Vaccines, Inc.

40 Landsdowne Street, Cambridge, MA 02139,

**USA** 

Trial Identifier: DEN-304

**IND Number:** 014292 **EudraCT Number:** Not available

Vaccine Names:

• Investigational vaccine: tetravalent dengue vaccine candidate (TDV)

comprised of a molecularly characterized, attenuated dengue serotype 2 strain (TDV-2), a dengue serotypes 2/1 chimeric strain (TDV-1), a dengue serotypes 2/3 chimeric strain (TDV-3), and a

dengue serotypes 2/4 chimeric strain (TDV-4).

• Placebo: saline solution.

**Date:** 29 October 2018

Version: Version 4.0

### 1.0 ADMINISTRATIVE INFORMATION

### 1.1 Contacts

| | Issue | Contact |
|---|---|---|
| | Serious adverse event and pregnancy reporting | PPD |
| | | Fax and telephone numbers for serious adverse event and pregnancy reporting will be provided to the site. |
| | Medical Monitor<br>(medical advice on conduct of protocol<br>or compound) | Emergency medical contact information will be provided to the site. |
| | Responsible Medical Officer<br>(carries overall responsibility for the<br>conduct of the trial) | Emergency medical contact information will be provided to the site. |
| | commerc | Jal Use omis |
| | Responsible Medical Officer (carries overall responsibility for the conduct of the trial) | |
| Property | | |

This trial will be conducted with the highest respect for the individual participants in accordance with the requirements of this clinical trial protocol and also in accordance with the following.

The ethical principles that have their origin in the Dool.

International C

- International Council for Harmonization of Technical Requirements for Pharmaceuticals E6 Good Clinical Practice: Consolidated Guideline.
- All applicable laws and regulations, including, but not limited to those related to data privacy and clinical trial disclosure.



### **INVESTIGATOR AGREEMENT**

I confirm that I have read and that I understand this protocol, the Investigator's Brochure, and any other product information provided by the Sponsor. I agree to conduct this trial in accordance with the requirements of this protocol and also protect the rights, safety, privacy, and well-being of trial subjects in accordance with the following:

- The ethical principles that have their origin in the Declaration of Helsinki.
- International Council for Harmonization of Technical Requirements for Pharmaceuticals, E6 Good Clinical Practice: Consolidated Guideline.
- All applicable laws and regulations, including, but not limited to those related to data privacy and clinical trial disclosure.
- Regulatory requirements for reporting serious adverse events defined in Section 10.4 of this protocol.
- Terms outlined in the Clinical Trial Site Agreement.
- Appendix A Responsibilities of the Investigator.

I further authorize that my personal information may be processed and transferred in accordance with the uses contemplated in Appendix B of this protocol.

| Signature of Investigator | Date |
|------------------------------------|------|
| Signature of Investigator | |
| Investigator Name (print or type) | |
| Forno | |
| Investigator's Title | |
| 1 step | |
| Location of Facility (City, State) | |
| O. | |
| Location of Facility (Country) | |

# 1.3 Protocol Amendment Summary of Changes

This document describes the changes in reference to the Protocol incorporating Amendment No. 2. The primary purpose of this amendment is to remove the planned Day 120 (Month 4 [M4]) interim analysis. Minor grammatical and editorial changes are included for clarification purposes only. Full details on changes of text are given in Section 1.3.2.

### 1.3.1 Amendment History

| Date | Amendment Number | Amendment Type | Region |
|-------------------|------------------|-----------------|--------|
| 26 September 2016 | Initial Protocol | Not applicable | Global |
| 21 July 2017 | 1 | Substantial | Global |
| 29 October 2018 | 2 | Non-substantial | Global |

### 1.3.2 Summary of Changes

Amendment to Protocol Version 3.0, 21 July 2017

### **Rationale for the Amendment:**

The rationale for removing the planned Day 120 (M4) interim analysis is that it is no longer required.

The removal of this interim analysis has no impact on the final statistical analyses planned for this study, the scientific value of the study, the study conduct, or the safety of subjects enrolled.

The administrative trial information has been updated and the reference list has been checked and updated as needed.

Details of the changes are outlined below. In this section only (ie, not in the protocol body) all new text is shown in bold italics and any redundant text is marked using strikethrough.

| Section | Description of change | |
|---|---|---|
| 1.1 | Serious adverse event and pregnancy reporting | PPD |
| | | Fax and telephone numbers for serious adverse event and pregnancy reporting will be provided to the site. |
| 1.1 | Medical Monitor | PPD |
| | (medical advice on conduct of protocol or compound) | |
| | | Emergency medical contact information will be provided to the site. |
| 1.1 | Responsible Medical Officer (carries overall responsibility for the conduct of the trial) | PPD |
| | 0,0 | Emergency medical contact information will be provided to the site. |
| 1.2 | PPD | PPD |
| 1.2 | PPD | PPD |
| 2.0, 13.2 | 120 (M4). This analysis will be performed by a safe a selected independent contract research organ assignment but will not be involved in subseque conduct of the trial, including those at Takeda, to individual vaccine assignment until unblinding and pay 270 [M9] follow up visit). No modification interim analysis. More details regarding the interior analyses are planned. | ity data is planned when all subjects have completed Day separate group of unblinded statisticians and programmers nization (CRO) who will have access to individual vaccine and trial conduct. The rest of the personnel involved in the he CRO, and the trial sites, will remain blinded to after trial completion (database lock for data through the a to the trial will be made based on the results of this arim analysis will be provided in the SAP. No interim |
| 6.2 | The rationale for the proposed trial is given in S analysis. | ection 4.2. Refer to Section 13.2 for the planned interim |

**S**tob

# **TABLE OF CONTENTS**

| 1.0 | ADM | INISTRATIVE INFORMATION | 2 |
|---|---|---|---|
| 1. | .1 Co | ontactsoproval | |
| 1. | 2 Ar | pproval | 3 |
| 1. | .3 Pr | oproval | 5 |
| | 1.3.1 | Amendment History | 5 |
| | 1.3.2 | Summary of Changes | 5 |
| 2.0 | TRIA | L SUMMARY | 11 |
| 2. | 1 Sc | hedule of Trial Procedures | 20 |
| 3.0 | TRIA | hedule of Trial Procedures L REFERENCE INFORMATION ial-Related Responsibilities gnatory Principal Investigator st of Abbreviations orporate Identification ODUCTION ackground attionale for the Proposed Trial | 22 |
| 3. | 1 Tr | ial-Related Responsibilities | 22 |
| 3. | 2 Si | gnatory Principal Investigator | 22 |
| 3. | .3 Li | st of Abbreviations | 23 |
| 3. | 4 Co | orporate Identification | 24 |
| 4.0 | INTR | ODUCTION | 25 |
| 4. | 1 Ba | ickground | 25 |
| 4. | 2 Ra | tionale for the Proposed Trial. | 26 |
| 5.0 | | L OBJECTIVES AND ENDPOINTS | |
| 5. | .1 Ot | ojectives | 28 |
| | 5.1.1 | Primary Objective | 28 |
| | 5.1.2 | | 28 |
| 5. | 2 Er | idpoints | |
| | 5.2.1 | Primary Endpoint | 28 |
| | 5.2.2 | Secondary Endpoints | 28 |
| 6.0 | TRIA | L DESIGN AND DESCRIPTION | 30 |
| 6. | | ial Design | 30 |
| 6. | 2 Ju | stification for Trial Design, Dose, and Endpoints | 32 |
| 6, | 3\ Dı | rration of Subject's Expected Participation in the Entire Trial | 32 |
| 6. | 4 Pr | emature Termination or Suspension of Trial or Investigational Site | 32 |
| 6. | 6.4.1 | Criteria for Premature Termination or Suspension of the Trial | 32 |
| <b>)</b> | 6.4.2 | Criteria for Premature Termination or Suspension of Investigational Sites | |
| | 6.4.3 | Procedures for Premature Termination or Suspension of the Trial or the | |
| | | Participation of Investigational Site(s) | |
| 7.0 | SELE | CTION AND DISCONTINUATION/WITHDRAWAL OF SUBJECTS | 34 |

| | 7.1 | Inc | elusion Criteria | 34 |
|---|---|---|---|---|
| | 7.2 | Ex | clusion Criteria | 34 |
| | 7.3 | Cr | iteria for Delay of Vaccination and/or Blood Sampling | 36 |
| | 7.4 | Cr | iteria for Early Trial Termination of a Subject | 37 |
| | 7.5 | - Cr | iteria for Premature Discontinuation of Trial Vaccine Application | - 38 |
| 8.0 | ) Cl | LINI | CAL TRIAL MATERIAL MANAGEMENT | 40 |
| | 8.1 | Tri | CAL TRIAL MATERIAL MANAGEMENT. al Vaccines and Materials Dosage Form, Packaging, and Labeling Storage Dose and Regimen | 40 |
| | 8. | 1.1 | Dosage Form, Packaging, and Labeling | 40 |
| | 8. | 1.2 | Storage | 40 |
| | 8. | 1.3 | Dose and Regimen | 41 |
| | 8.2 | | al Vaccine Assignment and Dispensing Procedures | 41 |
| | 8.3 | Ra | ndomization Code Creation and Storage al Vaccine Blind Maintenance blinding Procedure | 42 |
| | 8.4 | Tri | al Vaccine Blind Maintenance | 42 |
| | 8.5 | Un | blinding Procedure | 42 |
| | 8.6 | Ac | countability and Destruction of Sponsor-Supplied vaccines | 43 |
| 9.0 | ) TI | RIAI | al Procedures | 45 |
| | 9.1 | Tri | al Procedures | 45 |
| | 9. | 1.1 | Informed Consent Form | 45 |
| | 9. | 1.2 | Demographics, Medical History and Prior Medications | |
| | 9. | 1.3 | Documentation of Trial Entrance/Randomization | |
| | 9. | 1.4 | Physical Examination. | |
| | 9. | 1.5 | Vital Signs | 47 |
| | 9. | 1.6 | Immunogenicity Assessments | |
| | 9. | 1.7 | Safety Assessments | |
| | 9. | 1.8 | Contraception and Pregnancy Avoidance Procedure | |
| | | | Pregnancy | |
| | | N 1/2 | Documentation of Subjects who are not Randomized | |
| | 9.2 | , | onitoring Subject Compliance to TDV or Placebo Administration | |
| | 93 | | hedule of Observations and Procedures | |
| X | | 3.1 | Pre-Vaccination Procedures (Day 1 [M0] and Day 90 [M3]) | |
| 7 | | 3.2 | Vaccination Procedures (Day 1 [M0] and Day 90 [M3]) | |
| ) | | 3.3 | Post Vaccination Procedures (Day 1 [M0] and Day 90 [M3]) | 49 |
| | 9 | 3.4 | Clinic Visits after Vaccination (Day 30 [M1], Day 120 [M4], and Day 270 | Z 1 |
| | 0.7 | 2 5 | [M9]) | |
| | 9 | 3.5 | Final (End of Trial) Visit | 52 |

| | 9.3.6 | Post-Trial Care | 52 |
|---|---|---|---|
| 9.4 | Bio | ological Sample Retention and Destruction | 52 |
| 10.0 | | RSE EVENTS | |
| 10. | 1 De | finitions | 253 |
| | 10 1 1 | Adverse Events | 53 |
| | 10.1.2 | Solicited Adverse Events | 53 |
| | 10.1.3 | Medically Attended Adverse Events | 55 |
| | 10.1.4 | Serious Adverse Events | 55 |
| 10.2 | 2 Ca | Solicited Adverse Events Medically Attended Adverse Events Serious Adverse Events usality of Adverse Events Relationship to Trial Procedures | 55 |
| | 10.2.1 | Relationship to Trial Procedures | 55 |
| 10.3 | 3 Ad | ditional Points to Consider for Adverse Events | 56 |
| 10.4 | 4 Pro | Collection and Reporting of Adverse Events | 57 |
| | 10.4.1 | Collection and Reporting of Adverse Events | 57 |
| | 10.4.2 | Collection and Reporting of Solicited Adverse Events | 58 |
| | | Collection and Reporting of Medically Attended Adverse Events | |
| | 10.4.4 | Collection and Reporting of Serious Adverse Events. | 58 |
| 10. | 5 Fol | llow-up Procedures | . 59 |
| | 10.5.1 | Adverse Events | 59 |
| | | Serious Adverse Events | |
| | 10.5.3 | Safety Reporting to Investigators, Institutional Review Boards, and Regulatory | |
| | | Authorities. | 59 |
| 44.0 | | Post-Trial Events | |
| | | -SPECIFIC REQUIREMENT(S) | |
| 11. | | al-Specific Committees | |
| 10.0 | | Data Monitoring Committee | |
| | 4 | HANDLING AND RECORDKEEPING | |
| 12. | | ectronic CRFs (eCRF) | |
| | | cord Retention | |
| 13.0 | b | ISTICAL METHODS | |
| N | | atistical and Analytical Plans | |
| | | Analysis Sets Analysis of Demographics and Other Passline Characteristics | |
| , | | Analysis of Demographics and Other Baseline Characteristics | |
| | | Safety Analysis | |
| 13.2 | | erim Analysis and Criteria for Early Termination | |
| 1 | ا 1111 ك | ormir amaryoto and ormena for Darry Tornination | 03 |

| 13.3 D | etermination of Sample Size | 65 |
|---|---|---|
| 14.0 QUA | LITY CONTROL AND QUALITY ASSURANCE | 66 |
| 14.1 Tı | rial-Site Monitoring Visits | 66 |
| 14.2 Pr | otocol Deviations | 266 |
| 14.3 Q | uality Assurance Audits and Regulatory Agency Inspections | 66 |
| 15.0 ETHI | CAL ASPECTS OF THE TRIAL | 67 |
| 15.1 In | uality Assurance Audits and Regulatory Agency Inspections CAL ASPECTS OF THE TRIAL stitutional Review Board ubject Information, Informed Consent, and Subject Authorization ubject Confidentiality ublication, Disclosure, and Clinical Trial Registration Policy | 67 |
| 15.2 St | ubject Information, Informed Consent, and Subject Authorization | 68 |
| 15.3 St | ubject Confidentiality | 69 |
| 15.4 Pu | ublication, Disclosure, and Clinical Trial Registration Policy | 69 |
| 15.4.1 | Publication and Disclosure | 69 |
| 15.4.2 | Clinical Trial Registration | 69 |
| 15.4.3 | Clinical Trial Results Disclosure | 70 |
| 15.5 In | surance and Compensation for Injury | 70 |
| 16.0 REFE | RENCES | 71 |
| | 4.0 | |
| LIST OF IN | Publication and Disclosure Clinical Trial Registration Clinical Trial Registration Clinical Trial Results Disclosure surance and Compensation for Injury TEXT TABLES | |
| Table 8.a | Sponsor-Supplied Vaccines and Placebo | 41 |
| Table 10.a | Local and Systemic AEs. | |
| Table 10.b | Solicited Safety Parameters | |
| Table 16.a | Serology Plan | 79 |
| 10010 10.0 | Solotogy 1 Manual | |
| I ICT OF IN | -TEXT FIGURES | |
| | | 10 |
| Figure 2.a | Schematic of Trial Design | |
| Figure 6.a | Schematic of Trial Design | 31 |
| . 0 | | |
| LIST OF AF | PENDICES | |
| Appendix A | Responsibilities of the Investigator | 73 |
| Appendix B | Investigator Consent to Use of Personal Information | 75 |
| Appendix C | Elements of the Subject Informed Consent Form | |
| 40. | Serology Plan | 79 |

### 2.0 TRIAL SUMMARY

| Name of Sponsor: | | Product Name: |
|---|---|---|
| Takeda Vaccines, Inc | Takeda Vaccines, Inc Tetravalent Dengue Vaccine Candidate (TDV) | |
| 40 Landsdowne Street, Cambridge, MA | 40 Landsdowne Street, Cambridge, MA 02139, USA | |
| Trial Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Demonstrate Lot-to-Lot Consistency | | |
| of 3 Lots of a Tetravalent Dengue Vaccine Candidate in Healthy Adults in Non-Endemic Country(ies) for Dengue. | | |
| IND No.: 014292 EudraCT No.: Not applicable | | |
| Trial Identifier: DEN-304 Phase: 3 Trial Blinding Schema: Double-Blind | | |

### **Background and Rationale:**

Dengue fever is caused by infection with the wild type dengue virus (DENV), a ribonucleic acid virus that occurs as 4 recognized serotypes, DENV-1, DENV-2, DENV-3, or DENV-4. These dengue viruses are transmitted from human to human by mosquitoes (primarily *Aedes aegypti*). The 4 dengue viruses are endemic in Asia, Central and South America, the Caribbean, the Pacific Islands, and parts of Africa. There are an estimated 390 million dengue infections per year worldwide, which is more than 3 times the previous World Health Organization (WHO) estimate of 50 to 100 million cases. Every year, around 500,000 cases of dengue hemorrhagic fever (DHF) require hospitalization with an estimated death rate of 2.5%, primarily in children. It is estimated that 3.9 billion people are at risk of dengue infection.

Dengue fever is clinically defined as an acute febrile illness with 2 or more of the following manifestations: headache, retro-orbital pain, myalgia, arthralgia, rash, hemorrhagic manifestations, or leucopenia, and occurrence at the same location and time as other confirmed cases of dengue fever. The most severe forms of dengue infection – DHF and dengue shock syndrome (DSS) – are life threatening. Primary infection with any one of the 4 dengue serotypes is thought to result in life-long protection from re-infection by the same serotype, but does not protect against a secondary infection by one of the other 3 dengue serotypes and may lead to an increased risk of severe disease (DHF/DSS).

Treatment of dengue fever is based solely on signs and symptoms, with fluid replacement required for hemorrhagic or shock cases. An antiviral therapy for dengue virus infection is not available. Preventive measures that rely on mosquito control and individual protection are of limited efficacy, complex to implement and questionable in terms of cost-effectiveness. There is a great unmet global public health need for a safe and effective vaccine to reduce the morbidity and mortality associated with dengue disease. Vaccine development has focused on tetravalent vaccines that provide protection against all 4 dengue serotypes simultaneously since all 4 dengue serotypes commonly co-circulate in endemic areas. A first tetravalent dengue vaccine (CYD-TDV) has been recently approved in some countries in Asia and Latin America. However, the initial findings suggest an unfavorable risk-benefit profile for younger subjects with the approved vaccine. Additionally, vaccine efficacy was different between serotypes and depended on dengue pre-exposure status. Hence, there is a continued unmet public health need for safer and more efficacious dengue vaccines.

### Tetravalent Dengue Vaccine Candidate (TDV) - Background:

Takeda's TDV consists of 1 molecularly characterized, attenuated dengue serotype 2 virus strain and 3 chimeric recombinant dengue virus strains expressing surface antigens corresponding to dengue serotypes 1–4. The dengue serotype 2 strain (TDV-2) is based upon the attenuated laboratory-derived virus, DENV-2 Primary Dog Kidney (PDK)-53, originally isolated at Mahidol University, Bangkok, Thailand. The chimeric, attenuated vaccine strains for dengue serotypes 1, 3 and 4 were engineered by substituting the structural genes, pre-membrane (prM) and envelope (E), of TDV-2 with the prM and E genes of the wild type (DENV) virus strains, DENV-1 16007, DENV-3 16562 or DENV-4 1036 virus, respectively. Thus TDV is comprised of 4 dengue virus strains: a molecularly characterized, attenuated dengue serotype 2 strain (TDV-2), a dengue serotypes 2/1 chimeric strain (TDV-1), a dengue serotypes 2/3 chimeric strain (TDV-3), and a dengue serotypes 2/4 chimeric strain (TDV-4).

Nonclinical studies carried out in mice and nonhuman primates have demonstrated an acceptable safety, immunogenicity, and efficacy profile of Takeda's TDV. Additionally, data from completed phase 1 and phase 2

clinical trials in humans have shown satisfactory reactogenicity, safety and immunogenicity profiles of Takeda's TDV in healthy adults in non-endemic areas as well as in healthy adults and children in endemic areas in Asia and Latin America. Ongoing and completed phase 2 clinical trials have enabled the selection of a final TDV dose (lyophilized formulation) and a 2-dose vaccination regimen 3 months apart by subcutaneous (SC) injection for use in the pivotal program.

The current Investigator's Brochure contains additional product information and a more detailed review of pre-clinical and clinical trials.

### **Rationale for the Proposed Trial:**

Different production lots of TDV will be used in upcoming clinical trials. The WHO guidelines for independent lot release of vaccines specify that no new biological substance should be released until consistency of manufacturing and quality, as demonstrated by a consistent release of batches, has been established. In addition, the WHO recommends assessment of lot-to-lot consistency with the specific aim of comparing immunogenicity and safety between equal numbers of subjects who receive different lots. The primary objective of this trial is to investigate lot-to-lot consistency in terms of equivalence of the immune responses induced by 3 consecutive TDV lots in a healthy adult population in country(ies) non-endemic for dengue. It is anticipated that the conclusion from this trial can be extrapolated to age groups other than adults. This trial will also contribute to the safety database of dengue naive adult subjects included in the dengue clinical development program.

To minimize bias, the trial will be randomized, placebo-controlled, and double-blind. Subjects with a history of flavivirus infection or vaccination, or prolonged (≥1 year) habitation in a dengue endemic area will be excluded to minimize confounding factors. There will be 4 trial groups, 3 TDV groups and a placebo group. In each group, 2 doses of either TDV (Lots 1, 2, or 3) or placebo (0.9% saline) will be administered 3 months apart (ie, Day 1 [Month 0; M0] and Day 90 [Month 3; M3]).

Approximately 924 subjects are planned to be enrolled in the trial. Immunogenicity will be assessed in subjects included in the immunogenicity subset (TDV groups: 176 subjects each and placebo group: 88 subjects) and safety will be assessed in all subjects in each group (TDV groups: 264 subjects each and placebo group: 132 subjects). The immunogenicity assessment for the primary endpoint is planned at 1 month post second dose (Day 120 [M4]) to coincide with the anticipated peak in post-vaccination antibody titers. As the trial will be conducted in country(ies) non-endemic for dengue, 6 months follow-up duration after the last dose is considered adequate.

This trial will be conducted in accordance with the protocol, the International Council for Harmonization of Technical Requirements for Pharmaceuticals for Human Use and Good Clinical Practice (ICH-GCP) Guidelines and all applicable local laws and regulations, including, but not limited to those related to data privacy and clinical trial disclosure.

### **Trial Design:**

This is a randomized, double-blind, placebo-controlled phase 3 trial with 924 healthy subjects aged 18 to 60 years. The trial will be conducted in country(ies) non-endemic for dengue to investigate lot-to-lot consistency in terms of equivalence of the immunogenicity of 3 consecutive TDV lots administered as a 2-dose regimen 3 months apart via SC injection. Subjects will be randomized (2:2:2:1 ratio) to one of 4 trial groups to receive TDV (Lots 1, 2 or 3); 264 subjects per group) or placebo (132 subjects):

- Group 1: TDV Lot 1 administered on Day 1 (M0) and Day 90 (M3).
  - Group 2: TDV Lot 2 administered on Day 1 (M0) and Day 90 (M3).
- Group 3: TDV Lot 3 administered on Day 1 (M0) and Day 90 (M3).
- Group 4: Placebo administered on Day 1 (M0) and Day 90 (M3).

The sample size of 924 subjects (Groups 1-3: 264 subjects each and Group 4: 132 subjects) is intended to ensure sufficient size of the overall safety database in dengue non-endemic regions. A total of 616 subjects (Groups 1-3: 176 subjects each and Group 4: 88 subjects) is considered sufficient for immunogenicity assessments and is defined as the immunogenicity subset. Subjects will be randomly selected for inclusion in the immunogenicity subset using an interactive response technology (IRT).

All subjects will be followed-up for 6 months post second vaccination on Day 90 (M3) through Day 270 (M9), so the trial duration will be approximately 270 days (9 months) for each subject.

The schematic of the trial design is presented below in Figure 2.a.

Figure 2.a **Schematic of Trial Design** 



M=Month, V=Visit.

Note: Blood samples for immunogenicity will only be collected from the immunogenicity subset (Groups 1-3: 176 subjects each and Group 4: 88 subjects).

### Immunogenicity evaluation (immunogenicity subset):

Neutralizing antibodies (microneutralization test [MNT<sub>50</sub>]) will be measured using blood samples collected pre first vaccination (Day 1 [M0]) and post second vaccination (Day 120 [M4] and Day 270 [M9]).

### Safety evaluation (all subjects):

- Diary cards will be distributed for the recording of:
  - Solicited local adverse events (AEs) for 7 days following each TDV/placebo dose on Day 1 (M0) and Day 90 (M3) (day of vaccination + 6 days). These will include: injection site pain, injection site erythema, and injection site swelling.
  - Solicited systemic AEs for 14 days following each TDV/placebo dose on Day 1 (M0) and Day 90 (M3) (day of vaccination + 13 days). These will include: fever, headache, asthenia, malaise, and myalgia.
- Unsolicited AEs for 28 days following each TDV/placebo dose on Day 1 (M0) and Day 90 (M3) (day of vaccination + 27 days) will be collected by interview and recorded for all subjects.
- Serious adverse events (SAEs) and medically attended AEs (MAAEs) will be collected for the trial duration. MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria.

Data collection will be by electronic Case Report Form.

### **Primary Objective:**

• To demonstrate lot-to-lot consistency of 3 consecutive TDV lots in terms of equivalence of immune responses at 1 month post second dose.

### **Secondary Objectives:**

### Immunogenicity

- To describe the seropositivity rates for all dengue serotypes at 1 month and at 6 months post second TDV dose or placebo, where seropositivity is defined as a reciprocal neutralizing titer  $\ge 10$ .
- To describe the persistence of the immune response at 6 months post second dose of TDV or placebo in dengue-naive subjects.

### Safety

• To assess the safety profile following each vaccination or placebo in all groups.

# Subject Population: Healthy subjects: Yes Planned age: 18 to 60 years Planned number of subjects: 924

Planned number of groups: Three TDV groups (3 consecutive lots) and one placebo group in a 2:2:2:1 ratio

### **Criteria for Inclusion:**

- 1. The subject is aged 18 to 60 years, inclusive.
- 2. Individuals who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs), and the clinical judgment of the Investigator.
- 3. The subject signs and dates a written informed consent form and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements.
- 4. Individuals who can comply with trial procedures and are available for the duration of follow-up.

### **Criteria for Exclusion:**

- 1. Individuals with an elevated oral temperature ≥ 38°C (100.4°F) within 3 days of the intended date of vaccination (consider whether applicable as an exclusion criterion or criterion for delay, see below).
- 2. Known hypersensitivity or allergy to any of the vaccine components (including excipients of the investigational vaccines, control or placebo).
- 3. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the trial.
- Individuals with any history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (eg, Guillain-Barré syndrome).
- 5. Individuals with history or any illness that, in the opinion of the Investigator, might interfere with the results of the trial or pose additional risk to the subjects due to participation in the trial.
- 6. Known or suspected impairment/alteration of immune function, including:
  - a. Chronic use of oral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (M0) (use of inhaled, intranasal, or topical corticosteroids is allowed).
  - b. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥ 2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (M0).
  - c. Administration of immunoglobulins and/or any blood products within the 3 months prior to Day 1 (M0) or planned administration during the trial.
  - d. Receipt of immunostimulants within 60 days prior to Day 1 (M0).
  - e. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Day 1 (M0).
  - f. Human immunodeficiency virus (HIV) infection or HIV-related disease.
  - g. Hepatitis C virus infection.
  - h. Genetic immunodeficiency.
- 7. Abnormalities of splenic or thymic function.
- 8. Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
- 9. Individuals with any serious chronic or progressive disease according to judgment of the Investigator (eg, neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
- 10. Individuals with body mass index (BMI) greater than or equal to 35 kg/m2 (=weight in kg/[height in meters2]).
- 11. Individuals participating in any clinical trial with another investigational product 30 days prior to Day 1 (M0) or intent to participate in another clinical trial at any time during the conduct of this trial.
- 12. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or who are planning to receive any vaccine within 28 days of trial vaccine administration.
- 13. Individuals involved in the trial conduct or their first degree relatives.
- 14. Individuals with history of substance or alcohol abuse within the past 2 years.

- 15. Female subjects who are pregnant or breastfeeding.
- 16. Females of childbearing potential<sup>1</sup> who are sexually active, and who have not used any of the acceptable contraceptive methods<sup>2</sup> for at least 2 months prior to Day 1 (M0).
- 17. Females of childbearing potential who are sexually active, and who refuse to use an acceptable contraceptive method up to 6 weeks after the last dose of trial vaccine (Day 90 [M3]). In addition, they must be advised not to donate ova during this period.
- 18. Any positive or indeterminate pregnancy test.
- 19. Previous and planned vaccination (during the trial conduct), against any flavivirus including dengue, yellow fever (YF), Japanese encephalitis (JE) viruses or tick-borne encephalitis.
- 20. Previous participation in any clinical trial of a dengue or other flavivirus (eg, West Nile [WN] virus) candidate vaccine, except for subjects who received placebo in those trials.
- 21. Subjects with a current or previous infection with a flavivirus such as dengue, Zika, YF, JE, WN fever, tick-borne encephalitis or Murray Valley encephalitis and subjects with a history of prolonged (≥1 year) habitation in a dengue endemic area.

There may be instances when individuals meet all entry criteria except one that relates to transient clinical circumstances (e.g., body temperature elevation or recent use of excluded medication or vaccine[s]). Under these circumstances, eligibility for trial enrollment may be considered if the appropriate window for delay has passed, inclusion/exclusion criteria have been rechecked, and if the subject is confirmed to be eligible.

### Criteria for delay of vaccination at Day 90 (M3):

If any of the criteria below occur at the time scheduled for the trial vaccination at Day 90 (M3), the second dose may be administered at a later date as long as the subject is otherwise eligible to continue trial participation. In certain situations, the period of delay may lead to deviation from the time window for the second dose at Day 90 (M3). The decision to vaccinate in those situations will be made by the Investigator. The following clinical circumstances warrant a delay for administration of the vaccination at Day 90 (M3):

- 1. Individuals with a clinically significant active infection (as assessed by the Investigator) or temperature >38.0°C (>100.4°F) within 3 days of intended trial vaccination.
- 2. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to planned vaccination or blood sampling.
- 3. Known or suspected altered or impaired immune function as specified under the exclusion criteria.

### Criteria for contraindication to vaccination at Day 90 (M3):

There are also circumstances under which receipt of the second dose at Day 90 (M3) is contraindicated in this trial. These circumstances include but are not limited to anaphylaxis or severe hypersensitivity reactions following the first trial vaccination at Day 1 (M0). If these reactions occur, the subject must not receive the trial vaccination at Day 90

<sup>&</sup>lt;sup>1</sup> Defined as status post onset of menarche and not meeting any of the following conditions: bilateral tubal ligation (at least 1 year previously), bilateral oophorectomy (at least 1 year previously) or hysterectomy.

<sup>&</sup>lt;sup>2</sup> Hormonal contraceptives (e.g., oral, injection, transdermal patch, implant, cervical ring), barrier method (condom with spermicide or diaphragm with spermicide) each and every time during intercourse, intrauterine device (IUD), monogamous relationship with vasectomized partner (partner must have been vasectomized for at least 6 months prior to Day 1 [M0]). Other contraceptive methods may be considered in agreement with the Sponsor and will be approved by the appropriate ethics committee.

 29 October 2018

(M3) but will be encouraged to continue trial participation for safety follow-up.

### **Trial vaccines**

The investigational vaccine is TDV, a tetravalent dengue vaccine comprised of 1 molecularly characterized, attenuated dengue virus strain, and 3 chimeric dengue virus strains with

TDV-1, TDV-2, TDV-3, and TDV-4, respectively.

Placebo

Normal saline for injection (0.9% saline).

Route of administration

SC route

### **Duration of the Trial:**

The trial duration for each subject will be approximately 270 days (9 months).

### Period of Evaluation:

For the duration of a subject's participation.

### Main Criteria for Evaluation and Analyses:

### **Primary Endpoint:**

• Geometric mean titers (GMT) of neutralizing antibodies (by MNT<sub>50</sub>) for each of the 4 dengue serotypes at Day 120 (M4) in the immunogenicity subset.

### **Secondary Endpoints:**

Immunogenicity (immunogenicity subset)

Seropositivity rates (% of seropositive subjects) for each of the 4 dengue serotypes at Day 120 (M4) and Day 270 (M9).

Note: Seropositivity is defined as a reciprocal neutralizing titer  $\geq 10$ .

GMTs of neutralizing antibodies (by MNT<sub>50</sub>) for each of the 4 dengue serotypes at Day 270 (M9).

Safety (all subjects)

- Frequency and severity of solicited local (injection site) AEs for 7 days (day of vaccination + 6 days) and solicited systemic AEs for 14 days (day of vaccination + 13 days) after each TDV/placebo dose on Day 1 (M0) and Day 90 (M3).
- Percentage of subjects with any unsolicited AEs for 28 days (day of vaccination + 27 days) after TDV/placebo dose on Day 1 (M0) and Day 90 (M3).
- Percentage of subjects with SAEs throughout the trial.
- Percentage of subjects with MAAEs throughout the trial.

### **Statistical Considerations:**

### Analysis sets

Safety set: The safety set will consist of all subjects who received at least 1 dose of trial vaccine.

Full analysis set (FAS): The FAS will include all randomized subjects in the immunogenicity subset who received at least 1 dose of trial vaccine and for whom a valid pre-dose and at least one valid post-dose blood sample is taken.

Per–protocol set (PPS): The PPS will exclude all subjects seropositive for dengue virus at Baseline and will include all subjects in the FAS who have no major protocol violations. The major protocol violation criteria will be defined as part of the blinded data review prior to the unblinding of trial vaccine assignment. The categories of major protocol violations include: (1) not meeting selected entry criteria, (2) not receiving the correct randomly assigned trial vaccine or placebo, (3) receiving prohibited therapies, (4) not receiving 2 doses of trial vaccine or receiving the second trial dose inadmissibly outside of the visit window, and (5) other major protocol violations that may be identified during blinded data reviews.

All summaries and analyses of safety data will be based on subjects in the safety set. The primary immunogenicity

analyses will be based on the PPS; additional immunogenicity analyses may be provided based on the FAS.

### Analysis of demographics and other Baseline characteristics

Age, gender, race, and other Baseline characteristics will be summarized descriptively by trial group for all randomized subjects.

### Immunogenicity analysis (immunogenicity subset)

An immunogenicity subset of 616 subjects (TDV groups: 176 subjects each and placebo group: 88 subjects) will be randomly selected for the immunogenicity analyses (i.e., the immunogenicity subset).

For the primary and secondary immunogenicity endpoints (i.e., GMTs of neutralizing antibodies and seropositivity rates for each of the 4 dengue serotypes), descriptive statistics and 95% CIs will be provided by trial group for each applicable visit (Day 120 [M4] and Day 270 [M9]). Seropositivity is defined as a reciprocal neutralizing titer ≥10.

The primary endpoint will evaluate lot-to-lot consistency at Day 120 (M4). For each serotype, an analysis of variance (ANOVA) model on the natural logarithms of titers of dengue neutralizing antibodies will include data from the subjects in Groups 1-3 with trial group as a factor. A 95% CI will be provided for the 3 pairwise comparisons of log-transformed GMTs. The CIs will be back-transformed in order to report 95% CIs of the ratios in the original scale. For each pairwise comparison, equivalence of immune responses will be established if the 95% CI for the ratio is contained between equivalence margins of 0.5 and 2.0. Lot-to-lot consistency will be concluded if equivalence of immune responses is established for all pairwise comparisons and all 4 dengue serotypes. For the secondary endpoint of GMT at Day 270 (M9), a similar model will be fit.

For the secondary endpoint of seropositivity, 95% CIs for the difference in proportions between groups of interest for each dengue serotype at each applicable visit will be constructed using the Newcombe and Wilson method.

The primary immunogenicity analyses will be based on the PPS; other immunogenicity analyses may be provided based on the FAS.

### Safety analysis (all subjects)

All safety data will be summarized by trial group using the safety set.

### Solicited AEs

In all subjects, the presence and severity (Grade) of solicited local AEs (injection site pain, injection site erythema and injection site swelling) and solicited systemic AEs (fever, asthenia, malaise, headache and myalgia) will be collected for 7 days and 14 days, respectively, following each vaccination (including the day of vaccination) via collection of diary cards.

For each solicited AE, the number and percentage of subjects with local (injection site) and systemic AEs will be summarized by trial group and event severity for each day after each vaccination (ie, Day 1 through Day 7 for local [injection site] AEs and Day 1 through Day 14 for systemic AEs), and overall. Summaries of first onset of each event and the number of days subjects reported experiencing each event will also be provided. For subjects with more than 1 episode of the same event, the maximum severity will be used for tabulations.

Persistent/prolonged solicited local or systemic AEs continuing on Day 8 and Day 15, respectively, following each trial vaccination will be assessed separately. Unless otherwise specified these AEs will not be included in the analyses/tabulations of unsolicited AEs and will have separate listings.

### Unsolicited AEs

Unsolicited AEs will be assessed for 28 days following each TDV/placebo dose (day of vaccination + 27 days).

In all subjects, unsolicited AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) and summarized by System Organ Class (SOC) and Preferred Term (PT) for each trial group. AEs leading to trial or vaccine withdrawal will also be summarized for the duration of the trial.

Unsolicited AEs will be summarized as follows: by PT including events with frequency greater than a pre-defined frequency (the percentage will be specified in the statistical analysis plan); by SOC and PT; by SOC, PT, and severity; and by SOC, PT, and relationship to the investigational vaccine. Subjects reporting more than 1 occurrence for the

term (level) being summarized will be counted only once.

In all subjects, MAAEs will be collected throughout the trial. MAAEs will be coded using MedDRA, and summarized by SOC and PT for each trial group.

In all subjects, SAEs will be collected throughout the trial. SAEs will be coded using MedDRA, and summarized by SOC and PT for each trial group.

### **Sample Size Justification:**

It is assumed that the natural logarithms of titers of neutralizing antibodies for each of the 4 dengue serotypes are distributed as independent normal distributions, with standard deviations of 1.35, 0.86, 1.21, and 1.27, respectively. A sample size of 137 evaluable subjects in each of the 3 TDV groups (ie, Groups 1-3) is sufficient to achieve approximately 90% overall power for establishing lot-to-lot consistency in terms of equivalence of immune responses to 3 consecutive TDV lots based on the 95% CIs of the titer ratios, using equivalence margins of 0.5 and 2.0. This sample size assumes no variation among the 3 TDV lots; that is, for each serotype, the true ratio of GMT is 1.0 between the first and second lots and between the second and third lots.

Further adjusted for approximately 20% dropouts and non-evaluable subjects, the required sample size to evaluate lot-to-lot consistency is approximately 176 subjects for each TDV group (ie, Groups 1-3) and 88 subjects for the placebo group, given 2:2:2:1 randomization ratio between trial groups and taking into account ratio between the immunogenicity subset and its complement. Therefore, the immunogenicity subset will include 616 subjects.

To ensure sufficient size of the safety database in the dengue non-endemic regions, overall sample size for the trial is 924 subjects: 264 for each TDV group and 132 for placebo group.

### **Interim Analysis:**

No interim analyses are planned.

### **Data Monitoring Committee:**

A Data Monitoring Committee (DMC) will have oversight of this clinical trial. The DMC functions at a Takeda dengue program level and further information are available in the DMC Charter. Property of Takedai. For non-con

**DEN-304 Version 4.0 (29 October 2018)** 

 29 October 2018

| 2.1 | <b>Schedule</b> | of Trial | <b>Procedures</b> |
|-----|-----------------|----------|-------------------|

| Visit | 1 | 2 <sup>(a)</sup> | 3 | 4-(a) | 5 |
|---|---|---|---|---|---|
| Day | Day 1<br>M0 | Day 30<br>M1 | Day 90<br>M3 | Day 120<br>M4 | Day 270<br>M9 (ET) <sup>(b)</sup> |
| V'-'(1) | 11 | 30 days<br>(-1/+7) after | 90 days<br>(-4/+7) after | 30 days<br>(-1/+7) after | 180 days<br>(-7/+14) after |
| Visit window (days) | 1±n.a | Visit 1 | Visit 1 | Visit 3 | Visit 3 |
| Informed consent (c) | X | • | S | | |
| Assessment of eligibility criteria (d) | X | | | | |
| Demographics | X | | | | |
| Medical history | X | | | | |
| Concomitant medications/vaccinations (e) | X | X | X | X | X |
| Check contraindications to trial dose administration | X | | X | | |
| Check criteria for delay of trial dose administration | | 0/3 | X | | |
| Complete physical examination (f) | Χ ( | ), | X | | |
| Targeted physical examination (g) | <u>0</u> | X | | X | X |
| Vital signs <sup>(h)</sup> | X | X | X | X | X |
| Pregnancy test (i) | X | | X | | |
| Pregnancy avoidance guidance (i) | X<br>X<br>X | X | X | X | |
| Blood sample for dengue neutralizing antibodies (5 mL) (k) | OX. | | | X | X |
| Randomization | X | | | | |
| Trial vaccine administration (1) | X | | X | | |
| Injection site evaluation (m) | X | | X | | |
| Distribution | X | | X | | |
| Diary card Review/collection of solicited adverse events (n) | | X | | X | |
| Adverse events leading to withdrawal or discontinuation | X | X | X | X | X |
| Unsolicited adverse events (o) | X | X | X | X | |
| Serious adverse events (p) | X | X | X | X | X |
| Medically attended adverse events (p) | X | X | X | X | X |

ET=early termination, M=month, n.a=not applicable

<sup>(</sup>a) Visit 2 and Visit 4 should occur 30 days (at least 29 days) after the 1st and 2nd dose.

 29 October 2018

- (b) If the subject terminates early, Day 270 (M9) procedures should be performed.
- (c) Up to 28 days prior to the day of randomization.
- (d) Review of inclusion/exclusion criteria will be performed prior to administration of Dose 1 on Day 1 (M0). After eligibility is assessed and written informed consent has been obtained, subjects will be randomized to receive 2 doses of TDV or placebo by subcutaneous injection.
- (e) All medications and vaccine history from 1 month (minimum 28 days) prior to administration of each trial dose of TDV or placebo up to 1 month (minimum 28 days) thereafter, steroids and immunostimulants within 60 days prior to Day 1 (M0), immunoglobulins and blood products within 3 months prior to Day 1 (M0), and immunosuppressive therapy within 6 months prior to Day 1 (M0). Concomitant medication/vaccination will be collected throughout the trial conduct.
- (f) Physical examination including measurement of weight and height; body mass index (BMI) will be calculated. Measurement of height is only required at Day 1 (M0).
- (g) Subjects may undergo a brief symptom-directed physical examination. Clinically significant changes from the Baseline examination should be recorded in the subject's source documents and electronic Case Report Form (eCRF).
- (h) Vital signs including (but not limited to) the measurement of systolic blood pressure/diastolic blood pressure, heart rate, and body temperature.
- (i) Pregnancy testing (serum or urine) for females of childbearing potential. Results must be confirmed and documented as negative prior to each trial dose administration. Additional pregnancy tests may be performed during the trial if deemed necessary by the Investigator.
- (j) Females of childbearing potential who are sexually active will be reminded during trial visits to adhere to acceptable contraceptive methods up to 6 weeks post second trial vaccination at Day 90 (M3). Subjects will be provided with information on acceptable methods of contraception as part of the subject informed consent process and will be asked to sign a consent form stating that they understand the requirements for avoidance of pregnancy and donation of ova.
- (k) Blood samples for immunogenicity assessments for subjects included in the immunogenicity subset. The blood sample on Day 1 (M0) should be taken prior to administration of Dose 1. The blood sample on Day 120 (M4) should be taken at least 29 days (-1, 7 days) after administration of Dose 2. At Day 270 (M9) a final blood sample will be taken.
- (l) Subjects will be randomized to receive TDV (Lots 1, 2 or 3) or placebo.
- (m) Injection site pain, erythema, and swelling assessed by blinded trial staff for 30 minutes post-vaccination.
- (n) Review the diary card and collect solicited local adverse events (AEs) that occurred after vaccination:
  - 1) Solicited local (injection site) AE for 7 days following administration of each trial vaccination (day of vaccination + 6 days). If solicited local AEs continue on Day 8 following each trial vaccination, record the extended information on the Adverse Event eCRF.
  - 2) Solicited systemic AEs for 14 days following administration of each trial vaccination (day of vaccination + 13 days). The Investigator will categorize events by severity (mild, moderate or severe) and will assess causality to vaccine administration (related or not related). If solicited systemic AEs continue on Day 15 following each trial vaccination, record the extended information on the Adverse Event eCRF.
- (o) Unsolicited AEs for 28 days following each trial vaccination (day of vaccination + 27 days) will be collected by interview and recorded on Day 30 (M1) and Day 120 (M4). The Investigator will categorize events by severity (mild, moderate or severe) and will assess causality to trial dose administration (related or not related).
- (p) Medically attended AEs and serious AEs will be collected for the trial duration.

The Sponsor will perform all trial-related activities with the exception of those identified in the Trial-Related Responsibilities template. The identified vendors in the template for specific trial-related activities will perform these activities in full or in partners.

3.2 Signatory Principle.

The Sponsor will select a Signatory Principal Investigator from the Investigators who participate in the trial. Selection criteria for this Investigator will include significant knowledge of the trial Ape Trincip, agrees the agree of the and subject to the agree of the and subject to the agree of protocol, the investigational vaccine, their expertise in the therapeutic area and the conduct of clinical research as well as trial participation. The Signatory Principal Investigator will be required to review and sign the clinical trial report and by doing so agrees that it accurately describes the

to the applicable rems of Use Trial No. DEN-304  **Protocol Version 4.0** 

### 3.3 List of Abbreviations

Adverse Event AΕ **Body Mass Index** BMI

**CFR** Code of Federal Regulations **CSR** Clinical Study Report **DENV** Wild Type Dengue Virus

DENV-1, -2, -3, -4 Wild Type Dengue Virus Serotypes 1, 2, 3, and 4

Dengue Hemorrhagic Fever DHF **DMC** Data Monitoring Committee DSS Dengue Shock Syndrome

Е Envelope

eCRF electronic Case Report Form

FAS Full Analysis Set

Food and Drug Administration **FDA** Good Clinical Practice **GCP GMT** Geometric Mean Titer

International Council for Harmonization of Technical Requirements for Pharmaceuticals ICH

for Human Use

Inc Incorporated

IND Investigational New Drug **IRB** Institutional Review Board Interactive Response Technology **IRT** 

JΕ Japanese Encephalitis Month 0, 1, 3, 4, and 9 M0, -1, -3, -4, -9

MAAE Medically Attended Adverse Event

Medical Dictionary for Regulatory Activities MedDRA

Microneutralization Test 50%  $MNT_{50}$ 

Per-Protocol Set PPS prM pre-Membrane Preferred Term PT

Serious Adverse Event SAE Statistical Analysis Plan SAP

SC Subcutaneous SOC System Organ Class

**SUSAR** Suspected Unexpected Serious Adverse Reaction

**TDV** Tetravalent Dengue Vaccine Candidate TDV-4 Dengue Serotypes 2/4 Chimeric Strain TDV-1 Dengue Serotypes 2/1 Chimeric Strain TDV-3 Dengue Serotypes 2/3 Chimeric Strain

Molecularly Characterized, Attenuated Dengue Serotype 2 Strain

World Health Organization

West Nile Yellow Fever

Dengue fever is caused by infection with the wild type dengue virus (DENV), a ribonucleic acid virus that occurs as 4 recognized serotypes, DENV-1, DENV-2, DENV-3, or DENV-4. There dengue viruses are transmitted from human to human by mosquitoes (The 4 dengue viruses are endemic in Asia Collisions, and parts of Asia Collisions). Islands, and parts of Africa. There are an estimated 390 million dengue infections per year worldwide, which is more than 3 times the previous World Health Organization (WHO) estimate of 50 to 100 million cases. Every year, around 500,000 cases of dengue hemorrhagic fever (DHF) require hospitalization with an estimated death rate of 2.5%, primarily in children. It is estimated that 3.9 billion people are at risk of dengue infection [1-4].

Dengue fever is clinically defined as an acute febrile illness with 2 or more of the following manifestations: headache, retro-orbital pain, myalgia, arthralgia, rash, hemorrhagic manifestations, or leucopenia, and occurrence at the same location and time as other confirmed cases of dengue fever. The most severe forms of dengue infection – DHF and dengue shock syndrome (DSS) – are life threatening. Primary infection with any one of the 4 dengue serotypes is thought to result in life-long protection from re-infection by the same serotype, but does not protect against a secondary infection by one of the other 3 dengue serotypes and may lead to an increased risk of severe disease (DHF/DSS) [3-6].

Treatment of dengue fever is based solely on signs and symptoms, with fluid replacement required for hemorrhagic or shock cases. An antiviral therapy for dengue virus infection is not available. Preventive measures that rely on mosquito control and individual protection are of limited efficacy, complex to implement and questionable in terms of cost-effectiveness. There is a great, unmet global public health need for a safe and effective vaccine to reduce the morbidity and mortality associated with dengue disease [1-7]. Vaccine development has focused on tetravalent vaccines that provide protection against all 4 dengue serotypes simultaneously since all 4 dengue serotypes commonly co-circulate in endemic areas. A first tetravalent dengue vaccine (CYD-TDV) has been recently approved in some countries in Asia and Latin America [8]. However, the initial findings suggest an unfavorable risk-benefit profile for younger subjects with the approved vaccine. Additionally, vaccine efficacy was different between serotypes and depended on dengue pre-exposure status. Hence, there is a continued unmet public health need for safer and more efficacious dengue vaccines [9, 10].

### Tetravalent Dengue Vaccine Candidate (TDV) - Background:

Takeda's TDV consists of 1 molecularly characterized, attenuated dengue serotype 2 virus strain and 3 chimeric recombinant dengue virus strains expressing surface antigens corresponding to dengue serotypes 1–4. The dengue serotype 2 strain (TDV-2) is based upon the attenuated laboratory-derived virus, DENV-2 Primary Dog Kidney (PDK)-53, originally isolated at Mahidol University, Bangkok, Thailand [11]. The chimeric, attenuated vaccine strains for dengue serotypes 1, 3 and 4 were engineered by substituting the structural genes, pre-membrane (prM) and envelope (E), of TDV-2 with the prM and E genes of the wild type (DENV) virus strains, DENV-1 16007,

DENV-3 16562 or DENV-4 1036 virus, respectively [12]. Thus TDV is comprised of 4 dengue virus strains: a molecularly characterized, attenuated dengue serotype 2 strain (TDV-2), a dengue serotypes 2/1 chimeric strain (TDV-1), a dengue serotypes 2/3 chimeric strain (TDV-3), and a dengue serotypes 2/4 chimeric strain (TDV-4).

Nonclinical studies carried out in mice and nonhuman primates have demonstrated an acceptable safety, immunogenicity, and efficacy profile of Takeda's TDV. Additionally, data from completed phase 1 and phase 2 clinical trials in humans have shown satisfactory reactogenicity, safety and immunogenicity profiles of Takeda's TDV in healthy adults in non-endemic areas as well as in healthy adults and children in endemic areas in Asia and Latin America. Ongoing and completed phase 2 clinical trials have enabled the selection of a final TDV dose (lyophilized formulation) and a 2-dose vaccination regimen 3 months apart by subcutaneous (SC) injection for use in the pivotal program.

The current Investigator's Brochure contains additional product information and a more detailed review of pre-clinical and clinical trials [14].

### 4.2 Rationale for the Proposed Trial

Different production lots of TDV will be used in upcoming clinical trials. The WHO guidelines for independent lot release of vaccines specify that no new biological substance should be released until consistency of manufacturing and quality, as demonstrated by a consistent release of batches, has been established [14]. In addition, the WHO recommends assessment of lot-to-lot consistency with the specific aim of comparing immunogenicity and safety between equal numbers of subjects who receive different lots [15]. The primary objective of this trial is to investigate lot-to-lot consistency in terms of equivalence of the immune responses induced by 3 consecutive TDV lots in a healthy adult population in country(ies) non-endemic for dengue. It is anticipated that the conclusion from this trial can be extrapolated to age groups other than adults. This trial will also contribute to the safety database of dengue naive adult subjects included in the dengue clinical development program.

To minimize bias, the trial will be randomized, placebo-controlled and double-blind. Subjects with a history of flavivirus infection or vaccination, or prolonged (≥1 year) habitation in a dengue endemic area will be excluded to minimize confounding factors. There will be 4 trial groups, 3 TDV groups and a placebo group. In each group, 2 doses of either TDV (Lots 1, 2, or 3) or placebo (0.9% saline) will be administered 3 months apart (ie, Day 1 [Month 0; M0] and Day 90 [Month 3; M3]).

Approximately 924 subjects are planned to be enrolled in the trial. Immunogenicity will be assessed in subjects included in the immunogenicity subset (TDV groups: 176 subjects each and placebo group: 88 subjects) and safety will be assessed in all subjects in each group (TDV groups: 264 subjects each and placebo group: 132 subjects). The immunogenicity assessment for the primary endpoint is planned at 1 month post second dose (Day 120 [M4]) to coincide with the anticipated peak in post-vaccination antibody titers. As the trial will be conducted in region(s) non-endemic for dengue, 6 months follow-up duration after the last dose is considered adequate.

And a subject to the applicable of the properties of the propertie

### 5.0 TRIAL OBJECTIVES AND ENDPOINTS

### 5.1 Objectives

### 5.1.1 Primary Objective

• To demonstrate lot-to-lot consistency of 3 consecutive TDV lots in terms of equivalence of immune responses at 1 month post second dose.

### 5.1.2 Secondary Objectives

*Immunogenicity* 

- To describe the seropositivity rates for all dengue serotypes at 1 month and at 6 months post second TDV dose or placebo, where seropositivity is defined as a reciprocal neutralizing titer >10.
- To describe the persistence of the immune response at 6 months post second dose of TDV or placebo in dengue-naive subjects.

Safety

• To assess the safety profile following each vaccination or placebo in all groups.

### 5.2 Endpoints

### 5.2.1 Primary Endpoint

• Geometric mean titers (GMT) of neutralizing antibodies (by microneutralization test 50% [MNT<sub>50</sub>]) for each of the 4 dengue serotypes at Day 120 (M4) in the immunogenicity subset.

# 5.2.2 Secondary Endpoints

*Immunogenicity (immunogenicity subset)* 

• Seropositivity rates (% of seropositive subjects) for each of the 4 dengue serotypes at Day 120 (M4) and Day 270 (M9).

Note: Seropositivity is defined as a reciprocal neutralizing titer  $\geq 10$ .

• GMTs of neutralizing antibodies (by MNT<sub>50</sub>) for each of the 4 dengue serotypes at Day 270 (M9).

Safety (all subjects)

• Frequency and severity of solicited local (injection site) adverse events (AEs) for 7 days (day of vaccination + 6 days) and solicited systemic AEs for 14 days (day of vaccination + 13 days) after each TDV/placebo dose on Day 1 (M0) and Day 90 (M3).

ae trial.

ae trial.

ae trial.

ae trial.

Ays)

Ays)

April 2 applicable only and subject to the applicable only and applicable only applicable only and applicable only applicable on the applicable only applicable on the applicable only applicable only applicable only applicable only applicable only applicable on the applicable only applicable on the applicable only applicable on the applicable o

This is a randomized, double-blind, placebo-controlled phase 3 trial with 924 healthy subjects aged 18 to 60 years.

The trial will be conducted in country(ies) non-endemia for 1 consistency in terms of equivalence administration. administered as a 2-dose regimen 3 months apart via SC injection. Subjects will be randomized (2:2:2:1 ratio) to one of 4 trial groups to receive TDV (Lots 1, 2 or 3); 264 subjects per group) or placebo (132 subjects):

- Group 1: TDV Lot 1 administered on Day 1 (M0) and Day 90 (M3
- Group 2: TDV Lot 2 administered on Day 1 (M0) and Day 90 (M3).
- Group 3: TDV Lot 3 administered on Day 1 (M0) and Day 90 (M3).
- Group 4: Placebo administered on Day 1 (M0) and Day 90 (M3)

The sample size of 924 subjects (Groups 1-3: 264 subjects each and Group 4: 132 subjects) is intended to ensure sufficient size of the overall safety database in dengue non-endemic regions. A total of 616 subjects (Groups 1-3: 176 subjects each and Group 4: 88 subjects) is considered sufficient for immunogenicity assessments and is defined as the immunogenicity subset. Subjects will be randomly selected for inclusion in the immunogenicity subset using an interactive response technology (IRT).

All subjects will be followed-up for 6 months post second vaccination on Day 90 (M3) through Day 270 (M9), so the trial duration will be approximately 270 days (9 months) for each subject.

Hoperty of Lakedar For Hoper A schematic of the trial design is included as Figure 6.a. A schedule of trial procedures is provided

Figure 6.a **Schematic of Trial Design** 



M=Month, V=Visit.

Note: Blood samples for immunogenicity will only be collected from the immunogenicity subset (Groups 1-3: 176 subjects each and Group 4: 88 subjects).

### Immunogenicity evaluation (immunogenicity subset):

Neutralizing antibodies (MNT<sub>50</sub>) will be measured using blood samples collected pre first vaccination (Day 1 [M0]) and post second vaccination (Day 120 [M4] and Day 270 [M9]).

### Safety evaluation (all subjects):

- Diary cards will be distributed for the recording of:
  - Solicited local AEs for 7 days following each TDV/placebo dose on Day 1 (M0) and Day 90 (M3) (day of vaccination + 6 days). These will include: injection site pain, injection site erythema, and injection site swelling.
  - Solicited systemic AEs for 14 days following each TDV/placebo dose on Day 1 (M0) and Day 90 (M3) (day of vaccination + 13 days). These will include: fever, headache, asthenia, malaise, and myalgia.
- Unsolicited AEs for 28 days following each TDV/placebo dose on Day 1 (M0) and Day 90 (M3) (day of vaccination + 27 days) will be collected by interview and recorded for all subjects.

reins of Usi SAEs and MAAEs will be collected for the trial duration. MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria.

Data collection will be by electronic Case Report Form (eCRF).

### 6.2 Justification for Trial Design, Dose, and Endpoints

The trial design and the collection of solicited AEs, unsolicited AEs (non-serious AEs and SAEs), and MAAEs following trial dose administration are consistent with vaccine evaluation trials.

Ongoing and completed phase 2 trials have enabled the selection of a final TDV dose (lyophilized formulation) and a 2-dose vaccination regimen 3 months apart by SC injection for use in Takeda's pivotal dengue program.

The timing of the primary and secondary endpoints after vaccination is consistent with previous trials with TDV. Dengue neutralizing antibodies have been generally accepted as the immune response endpoint for dengue vaccine trials.

In order to maintain the double-blind design, a placebo (saline solution for injection) will be used in this trial. Enrollment into the 4 trial groups is unbalanced such that the group receiving TDV is over-represented.

As the trial will be conducted in areas non-endemic for dengue, a 6-month follow-up period after the second trial dose is considered adequate.

Justification of the sample size is included in Section 13.3.

The rationale for the proposed trial is given in Section 4.2.

### 6.3 Duration of Subject's Expected Participation in the Entire Trial

The trial duration for each subject will be approximately 270 days (9 months) including trial dose administration (Day 1 [M0] and Day 90 [M3]) and follow-up through Day 270 (M9).

### 6.4 Premature Termination or Suspension of Trial or Investigational Site

### Criteria for Premature Termination or Suspension of the Trial

The trial will be completed as planned unless one or more of the following criteria are satisfied that require temporary suspension or early termination of the trial.

- New information or other evaluation regarding the safety or efficacy of the investigational vaccine that indicates a change in the known risk/benefit profile, such that the risk/benefit is no longer acceptable for subjects participating in the trial.
- The Data Monitoring Committee (DMC) recommends that the trial should be suspended or terminated.

• Significant deviation from GCP that compromises the ability to achieve the primary trial objectives or compromises subject safety.

### 6.4.2 Criteria for Premature Termination or Suspension of Investigational Sites

A trial site may be terminated prematurely or suspended if the site (including the Investigator) is found in significant deviation from GCP, protocol, or contractual agreement, is unable to ensure adequate performance of the trial, or as otherwise permitted by the contractual agreement.

# 6.4.3 Procedures for Premature Termination or Suspension of the Trial or the Participation of Investigational Site(s)

In the event that the Sponsor, an institutional review board (IRB) or regulatory authority elects to e course of et al. For non commercial use only and sulfi terminate or suspend the trial or the participation of an investigational site, a trial-specific procedure for early termination or suspension will be provided by the Sponsor; the procedure will be followed by applicable investigational sites during the course of termination or trial suspension.

### 7.0 SELECTION AND DISCONTINUATION/WITHDRAWAL OF SUBJECTS

All entry criteria, including test results, need to be confirmed prior to randomization.

### 7.1 Inclusion Criteria

Subject eligibility is determined according to the following criteria:

- 1. The subject is aged 18 to 60 years, inclusive.
- 2. Individuals who are in good health at the time of entry into the trial as determined by medical history, physical examination (including vital signs) and the clinical judgment of the Investigator.
- 3. The subject signs and dates a written informed consent form and any required privacy authorization prior to the initiation of any trial procedures, after the nature of the trial has been explained according to local regulatory requirements (Appendix C).
- 4. Individuals who can comply with trial procedures and are available for the duration of follow-up.

### 7.2 Exclusion Criteria

Any subject who meets any of the following criteria will not qualify for entry into the trial:

- 1. Individuals with an elevated oral temperature (≥38°C or 100.4°F) within 3 days of the intended date of vaccination (consider whether applicable as an exclusion criterion or criterion for delay, see Section 7.3).
- 2. Known hypersensitivity or allergy to any of the vaccine components (including excipients of the investigational vaccine or placebo).
- 3. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the trial.
- 4. Individuals with any history of progressive or severe neurologic disorder, seizure disorder or neuro-inflammatory disease (eg, Guillain-Barré syndrome).
- 5. Individuals with history or any illness that, in the opinion of the Investigator, might interfere with the results of the trial or pose additional risk to the subjects due to participation in the trial.
- 6. Known or suspected impairment/alteration of immune function, including:
  - a. Chronic use of oral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (M0) (use of inhaled, intranasal, or topical corticosteroids is allowed).
  - b. Receipt of parenteral steroids (equivalent to 20 mg/day prednisone ≥12 weeks/≥ 2 mg/kg body weight/day prednisone ≥2 weeks) within 60 days prior to Day 1 (M0).
  - c. Administration of immunoglobulins and/or any blood products within the 3 months prior to Day 1 (M0) or planned administration during the trial.

- d. Receipt of immunostimulants within 60 days prior to Day 1 (M0).
- in of Use e. Immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within 6 months prior to Day 1 (M0).
- f. Human immunodeficiency virus (HIV) infection or HIV-related disease.
- g. Hepatitis C virus infection.
- h. Genetic immunodeficiency.
- 7. Abnormalities of splenic or thymic function.
- 8. Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
- 9. Individuals with any serious chronic or progressive disease according to judgment of the Investigator (eg, neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease).
- 10. Individuals with body mass index (BMI) greater than or equal to 35 kg/m<sup>2</sup> (= weight in kg/[height in meters<sup>2</sup>]).
- 11. Individuals participating in any clinical trial with another investigational product 30 days prior to Day 1 (M0) or intent to participate in another clinical trial at any time during the conduct of this trial.
- 12. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or who are planning to receive any vaccine within 28 days of trial vaccine administration.
- 13. Individuals involved in the trial conduct or their first degree relatives.
- 14. Individuals with history of substance or alcohol abuse within the past 2 years.
- 15. Female subjects who are pregnant or breastfeeding.
- 16. Females of childbearing potential who are sexually active, and who have not used any of the acceptable contraceptive methods for at least 2 months prior to Day 1 (M0).
  - a. Of childbearing potential is defined as status post onset of menarche and not meeting any of the following conditions: bilateral tubal ligation (at least 1 year previously), bilateral oophorectomy (at least 1 year previously) or hysterectomy.
  - b. Acceptable birth control methods are defined as one or more of the following:
    - Hormonal contraceptive (such as oral, injection, transdermal patch, implant, cervical ring).
    - Barrier method (condom with spermicide or diaphragm with spermicide) each and every time during intercourse.
    - Intrauterine device (IUD). iii.
    - Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least 6 months prior to Day 1 (M0).
Other contraceptive methods may be considered in agreement with the Sponsor and will be approved by the appropriate ethics committee.

- 17. Females of childbearing potential who are sexually active, and who refuse to use an acceptable contraceptive method up to 6 weeks after the last dose of trial vaccine (Day 90 [M3]). In addition, they must be advised not to donate ova during this period (Section 9.1.9).
- 18. Any positive or indeterminate pregnancy test.
- 19. Previous and planned vaccination (during the trial conduct) against any flavivirus including dengue, yellow fever (YF), Japanese encephalitis (JE) viruses or tick-borne encephalitis.
- 20. Previous participation in any clinical trial of a dengue or other flavivirus (eg, West Nile [WN] virus) candidate vaccine, except for subjects who received placebo in those trials.
- 21. Subjects with a current or previous infection with a flavivirus such as dengue, Zika, YF, JE, WN fever, tick-borne encephalitis or Murray Valley encephalitis and subjects with a history of prolonged (≥1 year) habitation in a dengue endemic area.

There may be instances when individuals meet all entry criteria except one that relates to transient clinical circumstances (eg, body temperature elevation or recent use of excluded medication or vaccine[s]). Under these circumstances, eligibility for trial enrollment may be considered if the appropriate window for delay has passed, inclusion/exclusion criteria have been rechecked, and if the subject is confirmed to be eligible.

# 7.3 Criteria for Delay of Vaccination and/or Blood Sampling

After enrollment, subjects may encounter clinical circumstances that warrant a delay in the administration of trial vaccination. These situations are listed below. In the event that a subject meets a criterion for delay of vaccination, the subject may receive trial vaccination once the window for delay has passed as long as the subject is otherwise eligible for trial participation.

If any of the criteria below occur at the time scheduled for the trial vaccination at Day 90 (M3), the second dose may be administered at a later date as long as the subject is otherwise eligible to continue trial participation. In certain situations, the period of delay may lead to deviation from the time window for the second dose at Day 90 (M3). The decision to vaccinate in those situations will be made by the Investigator. The following clinical circumstances warrant a delay for administration of the vaccination at Day 90 (M3):

- 1. Individuals with a clinically significant active infection (as assessed by the Investigator) or temperature >38.0°C (>100.4°F) within 3 days of intended trial vaccination (see Section 7.2).
- 2. Individuals who received any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to planned vaccination or blood sampling.
- 3. Known or suspected altered or impaired immune function as specified under the exclusion criteria (see Section 7.2).

# Criteria for contraindication to vaccination at Day 90 (M3):

There are also circumstances under which receipt of the second dose at Day 90 (M3) is contraindicated in this trial. These circumstances include but are not limited to anaphylaxis or severe hypersensitivity reactions following the first trial vaccination at Day 1 (M0). If these reactions occur, the subject must not receive the trial vaccination at Day 90 (M3) but will be encouraged to continue trial participation for safety follow-up.

#### 7.4 Criteria for Early Trial Termination of a Subject

Under some circumstances, a subject's trial participation may be terminated early. This means that no further trial procedures (including data collection) will be performed on that subject beyond the specific date of early termination. The primary reason for early termination of the subject from the trial should be recorded in the eCRF "end of trial visit" page using the following categories. For screen failure subjects, refer to Section 9.1.10.

- 1. Adverse Event: The subject has experienced an AE (irrespective of being related/unrelated to the trial vaccine or trial-related procedures) that requires early termination because continued participation imposes an unacceptable risk to the subject's health and/or the subject is unwilling to continue participation because of the AE. If the subject is unwilling to continue because of the AE the primary reason for early termination in this case will be 'withdrawal due to AE' and not 'withdrawal of consent', see below. Any ongoing AEs leading to early termination should be followed by the Investigator until resolution or stabilization.
- 2. Lost to follow-up: The subject did not return to the clinic and at least three attempts to contact the subject were unsuccessful. Attempts to contact the subject must be documented.
- 3. Withdrawal of consent: The subject wishes to withdraw from the trial. The primary reason for early termination will be 'withdrawal of consent' if the subject withdraws from participation due to a non-medical reason (ie, reason other than AE). The reason for withdrawal, if provided, should be recorded in the eCRF.
  - Note: All attempts should be made to determine the underlying reason for the withdrawal and, where possible, the primary underlying reason should be recorded.
- 4. Premature trial termination by Sponsor, a regulatory agency, the IRB, or any other authority. If the clinical trial is prematurely terminated by the Sponsor, the Investigator is to promptly inform the trial subjects and local IRB and should assure appropriate follow-up for the subjects. The primary reason for early termination in this case will be 'trial termination'.
- Subject's death during trial participation. Subject 6. Other.

Note: The specific reasons should be recorded in the "specify" field of the eCRF.

# 7.5 Criteria for Premature Discontinuation of Trial Vaccine Application

Early trial termination of a subject will by default prevent the subject from continued trial vaccine application as the subject will no longer be participating in the trial. In addition to early termination criteria (see Section 7.4), other situations may apply in which subjects may continue participating in the trial (eg, contributing safety data according to protocol) but trial vaccine application is discontinued selectively. Regardless of the reasons for the discontinuation of trial vaccine application, this must be documented as a protocol deviation. Even if the subject is deemed ineligible to receive trial vaccine, all efforts should be made to continue the collection of safety data according to protocol. In addition, the primary reason for premature discontinuation of trial vaccine application should be recorded in the eCRF, "end of trial vaccine application" page using the following categories:

- 1. Adverse Event: The subject has experienced an AE (irrespective of being related/unrelated to the trial vaccine or trial-related procedures) for which subsequent trial vaccine applications impose an unacceptable risk to the subject's health, but the subject may continue trial participation for safety, or a subset of other trial procedures.
- 2. Lost to follow-up: The subject did not return to the clinic and at least three attempts to contact the subject were unsuccessful. Attempts to contact the subject must be documented.
- 3. Withdrawal of consent: The subject wishes to withdraw from the trial. The primary reason for early termination will be 'withdrawal of consent" if the subject withdraws from participation due to a non-medical reason (ie, reason other than AE). The reason for withdrawal, if provided, should be recorded in the eCRF.
- 4. Premature trial termination by the Sponsor, a regulatory agency, the IRB, or any other authority.
  - If the clinical trial is prematurely terminated by the Sponsor, the Investigator is to promptly inform the trial subjects and local IRB and should assure appropriate follow-up for the subjects. The primary reason for early termination in this case will be 'trial termination'.
- 5. Subject's death during trial participation.
- 6. Protocol deviation: A protocol deviation is any change, divergence, or departure from the trial design or procedures of a trial protocol. The subject may remain in the trial unless continuation in the trial jeopardizes the subject's health, safety or rights (see Section 7.4).
- 7. Pregnancy: Any subject who, despite the requirement for adequate contraception, becomes pregnant during the trial will not receive further trial vaccine applications. Pregnant subjects should, however, be asked to continue participating in the trial contributing data to the safety follow-up according to protocol. In addition, the site should maintain contact with the pregnant subject and complete a "Clinical Trial Pregnancy Form" as soon as possible. The subject should be followed-up until the birth of the child, or spontaneous or voluntary termination; when pregnancy outcome information becomes available, the information should be captured

ARF. Terrison of the applicable to noncommercial use only and subject to the applicable. For noncommercial use only and subject to the applicable.

## 8.0 CLINICAL TRIAL MATERIAL MANAGEMENT

This section contains information regarding all vaccines and materials provided directly by the Sponsor, and/or sourced by other means, that are required by the trial protocol, including important sections describing the management of clinical trial material.

## 8.1 Trial Vaccines and Materials

The investigational vaccine is TDV, a tetravalent dengue vaccine comprised of 1 molecularly characterized, attenuated dengue virus strain, and 3 chimeric dengue virus strains

TDV-1, TDV-2,

TDV-3, and TDV-4, respectively.

Placebo is a normal saline solution (0.9% NaCl) for injection.

# 8.1.1 Dosage Form, Packaging, and Labeling

# TDV Kits (TDV and TDV diluent):

Manufacturing of monovalent bulk vaccine substances of TDV, mixing of the four TDV vaccine substances, filling into vials, and lyophilization of TDV is done at

Lyophilized TDV is presented in a single-dose CCI

TDV diluent (37 mM sodium chloride solution) is manufactured by

. CCI

TDV and TDV diluent vials are packaged together into single dose dispensing cartons. The vials will be labeled to contain pertinent trial information in local languages.

# Placebo:

Commercially available normal saline for injection (0.9% sodium chloride solution) will be used as placebo. The placebo is presented as single dose units for 0.5 mL dosing.

The Sponsor will supply study sites with TDV, TDV diluent and placebo packaged into single dose dispensing cartons. The vials and cartons will be labeled in a blinded fashion that will contain pertinent trial information in local languages. Further details can be found in the Pharmacy Manual.

# 8.1.2 Storage

The trial vaccines (TDV and placebo) and TDV diluent will be shipped in refrigerated containers at 2°C to 8°C. From receipt and prior to use, trial vaccines and TDV diluent must be protected from light and stored at 2°C to 8°C in a refrigerator, do not freeze.

All clinical trial material must be kept in an appropriate, limited-access, secure place until it is used or returned to the Sponsor or designee for destruction. All Sponsor-supplied vaccines must be stored under the conditions specified on the label, and remain in the original container until dispensed. A daily temperature log of the vaccine storage area must be maintained every working day. Temperature excursions must be reported to the Sponsor as soon as possible and use of these vaccines and TDV diluent requires Sponsor approval.

# 8.1.3 Dose and Regimen

Trial vaccine doses that will be provided to each trial group are presented in Table 8.a.

The 0.5 mL trial vaccine doses will be prepared and administered by the unblinded pharmacist or vaccine administrator according to the instructions in the Pharmacy Manual or per Sponsor instructions.

TDV and placebo will be administered by the SC route.

Table 8.a Sponsor-Supplied Vaccines and Placebo

| Group | Number of subjects | Day 1 (M0) | Day 90 (M3) |
|---------|--------------------|---------------|---------------|
| Group 1 | 264 | TDV lot 1, SC | TDV lot 1, SC |
| Group 2 | 264 | TDV lot 2, SC | TDV lot 2, SC |
| Group 3 | 264 | TDV lot 3, SC | TDV lot 3, SC |
| Group 4 | 132 | Placebo, SC | Placebo, SC |

M=Month, SC=subcutaneous

# 8.2 Trial Vaccine Assignment and Dispensing Procedures

The vaccine to be used will be identifiable by a unique identification number and managed by IRT. Refer to Section 8.6 for accountability of Sponsor-supplied vaccines.

The Investigator or designee will use IRT at subject enrollment to obtain the subject number. This number will be used throughout the trial.

The Investigator or designee will use IRT on the day of first dosing (Day1 [M0]) to provide the necessary subject identifying information.

The Investigator or designee will use IRT at each dispensing visit to obtain the vaccination identification number for the vaccine dose.

The Investigator or designee will be responsible for overseeing the administration of vaccine to subjects enrolled in the trial according to the procedures stipulated in this trial protocol. The vaccine will be administered only by unblinded personnel who are qualified to perform that function under applicable laws and regulations for that specific trial.

• If Sponsor-supplied vaccine is lost or damaged, the site can request a replacement. Expired vaccines must not be administered.

Prior to vaccination, a subject must be determined to be eligible for trial vaccination and it must be clinically appropriate in the judgment of the Investigator to vaccinate. Eligibility for vaccination prior to first trial vaccine administration is determined by evaluating the entry criteria outlined in this protocol (Section 7.1 and Section 7.2).

Eligibility for subsequent trial vaccination is determined by the criteria outlined in Section 7.3

Trial vaccines should not be administered to individuals with known hypersensitivity to any component of the vaccines.

Standard immunization practices are to be observed and care should be taken to administer the injection by the SC route. In addition, the WHO recommendations to reduce anxiety and pain at the time of vaccination should be followed [16]. Before administering the vaccine, the vaccination site is to be disinfected with a skin disinfectant (eg, 70% alcohol). Allow the skin to dry. DO NOT inject intravascularly.

As with all injectable vaccines, trained medical personnel and appropriate medical treatment should be readily available in case of anaphylactic reactions following vaccination. For example, epinephrine 1:1000, diphenhydramine, and/or other medications for treating anaphylaxis should be available. These rescue medications will not be supplied by the Sponsor.

# 8.3 Randomization Code Creation and Storage

Randomization personnel of the Sponsor or designee will generate the randomization schedule(s). Randomization information will be stored in a secured area, accessible only by authorized personnel.

# **8.4** Trial Vaccine Blind Maintenance

The trial will be conducted in a double-blind manner meaning that the subject, those responsible for the evaluation of any trial endpoint and the Sponsor will be all unaware of which trial vaccine was administered. The investigational vaccine blind will be maintained using IRT. The subjects, data collectors (eg, Investigator), and data evaluators (eg, trial statisticians) are blinded. One or more designated pharmacist's/vaccine administrators at the site will be unblinded. These unblinded personnel will be responsible for receiving and storing the trial vaccines to ensure that the trial blind is not broken. They will also be responsible for the trial vaccine accountability. The unblinded personnel will have no role in data collection or evaluation.

# 8.5 Unblinding Procedure

The trial vaccine blind shall not be broken by the Investigator unless information concerning the trial vaccine is necessary for the medical treatment of the subject or is requested by the subject in case of pregnancy. In the event of a pregnancy or medical emergency, if possible, the medical monitor should be contacted before the trial vaccine blind is broken to discuss the need for unblinding.

For unblinding a subject, the trial vaccine blind can be obtained by the Investigator, by accessing the IRT.

The Sponsor's Pharmacovigilance Department must be notified as soon as possible if the trial vaccine blind is broken by the Investigator and the completed SAE or pregnancy form must be sent within 24 hours. The date, time, and reason the blind is broken must be recorded in the source document and the same information (except the time) must be recorded on the eCRF.

If any subject is unblinded, no further doses of trial vaccine are to be administered and the subject can remain in the trial for safety follow-up.

# 8.6 Accountability and Destruction of Sponsor-Supplied Vaccines

Vaccine supplies will be counted and reconciled at the site before being locally destroyed or returned to the Sponsor or designee as noted below. Sites will maintain source documents in addition to entering data in IRT.

The Investigator or designee must ensure that the Sponsor-supplied vaccines (including TDV diluent) are used in accordance with the approved protocol and are administered only to subjects enrolled in the trial. To document appropriate use of Sponsor-supplied vaccines (TDV and placebo), the Investigator must maintain records of all Sponsor-supplied vaccines (including TDV diluent) delivery to the site, site inventory, administration and use by each subject, and return to the Sponsor or designee.

Upon receipt of Sponsor-supplied vaccines, the Investigator or designee must verify the contents of the shipments against the packing list. The verifier should ensure that the quantity is correct, the trial vaccines are received within the labeled storage conditions (ie, no cold chain break has occurred during transit), and are in good condition. If quantity and conditions are acceptable, the Investigator or designee will acknowledge receipt of the shipment by recording in the IRT.

If there are any discrepancies between the packing list and the actual product received, the Sponsor or designee must be contacted to resolve the issue. The packing list should be filed in the Investigator's essential document file by a qualified Investigator designee.

The pharmacist (or designated individual) at each site must maintain 100% accountability for all Sponsor-supplied vaccines (including TDV diluent) received and administered during their entire participation in the trial. Proper vaccine accountability includes, but is not limited to:

- Verifying that the actual inventory matches the documented inventory.
- Verifying that the log is completed for the vaccine lot number used to prepare each dose.
- Verifying that all containers used are documented accurately on the log.
- Verifying that required fields are completed accurately and legibly.

If any dispensing errors or discrepancies are discovered, the Sponsor must be notified immediately.

The pharmacist (or designated individual) at each site must record the current inventory of all Sponsor-supplied vaccines (TDV and placebo) including TDV diluent on a Sponsor-approved vaccine accountability log. The following information will be recorded at a minimum: protocol number and title, name of Investigator, site identifier and number, description of Sponsor-supplied vaccines, expiry date and amount. The log (IRT) should include all required information as a separate entry for each subject to whom Sponsor-supplied vaccine is administered.

Prior to site closure or at appropriate intervals throughout the trial, before any clinical trial materials are returned to the Sponsor or designee for destruction, a representative from the Sponsor or designee will perform clinical trial material accountability and reconciliation. The Investigator will retain a copy of the documentation regarding clinical trial material accountability, return, and/or destruction, and originals will be sent to the Sponsor or designee.

The pharmacist (or designated individual) at each site will be responsible for vaccine accountability and will document receipt, use, return, or destruction of trial vaccines (TDV and placebo) including TDV diluent.

ewed by and luse only and luse only and property of Takeda. For non-commercial use only and property of Takeda. Vaccine accountability documentation will be reviewed by the unblinded monitor during clinical

The following sections describe the trial procedures and data to be collected. For each procedure, subjects are to be assessed by the same Investigator or site personnel whenever possible The Schedule of Trial Procedures is located in Section 2.1.

9.1.1 Informed Can

The requirements of the informed consent form are described in Section 15.2.

Informed consent must be obtained prior to the subject entering into the trial (up to 28 days prior to first administration of the trial vaccine), and before any protocol-directed procedures are performed.

A unique subject number will be assigned to each subject after informed consent is obtained from the IRT. If all eligibility criteria are fulfilled, this subject number will be used throughout the trial. Subject numbers assigned to subjects who fail screening should not be reused (see Section 9.1.10).

# 9.1.2 Demographics, Medical History and Prior Medications

Demographic information to be obtained will include age, sex, race and ethnicity as described by the subject.

Medical history will also be collected, including but not limited to any medical history that may be relevant to subject eligibility for trial participation such as prior vaccinations, concomitant medications, and previous and ongoing illnesses or injuries. Relevant medical history can also include any medical history that contributes to the understanding of an AE that occurs during trial participation, if it represents an exacerbation of an underlying disease/preexisting problem.

All medications and vaccine history from 1 month (minimum 28 days) prior to administration of each trial vaccine dose up to 1 month (minimum 28 days) thereafter, steroids and immunostimulants within 60 days prior to Day 1 (M0), immunoglobulins and blood products within 3 months prior to Day 1 (M0), and immunosuppressive therapy within 6 months prior to Day 1 (M0). Concomitant medication/vaccination will be collected throughout the trial conduct and are to be recorded on the "Medication History/Concomitant Medications" eCRF and in the subject's source document. The use of antipyretics and/or analgesic medications within 24 hours prior to vaccination must be identified and the reason for their use (prophylaxis versus treatment) must be described in the source documents or the eCRF. Medications taken for prophylaxis are those intended to prevent the onset of AEs following vaccination. Medications taken for treatment are intended to reduce or eliminate the presence of symptoms that are present. Trial vaccination should be delayed if subjects have used antipyretics and/or analgesic medication within 24 hours prior to vaccine administration.

Prohibited Therapies (Refer to Section 7.2):

- Parenteral immunoglobulin preparation, blood products, and/or blood-derived products within the 3 months prior to Day 1 (M0).
- Immunosuppressive therapy within 6 months or systemic (eg, oral or parenteral) corticosteroid treatment within 60 days prior to Day 1 (M0) or immunostimulants within 60 days prior to Day 1 (M0).
- Any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to Day 1 (M0) and Day 90 (M3), and 28 days after each trial vaccination.
- Any other dengue vaccines (investigational or licensed) for the entire trial period.
- Receipt of any other clinical trial product within 30 days prior to Day 1 (M0).

These data must be written in the source documents.

Medical history (including corresponding medication) to be obtained will include any significant conditions or diseases that have disappeared or resolved at or prior to signing of informed consent form.

## 9.1.3 Documentation of Trial Entrance/Randomization

Only subjects who have a signed informed consent form, meet all of the inclusion criteria and none of the exclusion criteria are eligible for entrance/randomization into the vaccination phase. The randomization schedule will be created and controlled by the IRT provider. The randomization specification will be approved by the Sponsor's trial statistician or designee.

If the subject is found to be ineligible for the randomization/trial phase, the Investigator should record the primary reason for screen failure on the subject enrollment log.

Subjects included in the immunogenicity subset will be randomly selected using IRT.

## 9.1.4 Physical Examination

Physical examinations must be performed by a qualified health professional in accordance with local regulations and licensing requirements and as designated on the Site Responsibility Delegation Log. A complete physical examination will be performed on Day 1 (M0) and Day 90 (M3) according to the Investigator's standard practice. A complete physical examination includes but is not limited to: auscultation of heart and lungs, palpation of the abdomen, inspection of extremities (including skin over intended vaccination site[s]), and a check of general appearance and the measurement of weight and height. BMI will be calculated. Height will be only measured on Day 1 (M0).

Additional physical examinations may be performed if indicated by a review of the subject's medical history. The findings should be documented in the subject's source document.

Targeted physical examination including but not limited to measurement of vital signs (see Section 9.1.5) will be performed at Day 30 (Month 1 [M1]), Day 120 (M4), and Day 270 (M9).

Clinically significant changes from the Baseline assessment must be recorded in the subject's source documents and the eCRF.

Symptom-directed physical examinations may be performed if deemed necessary.

# 9.1.5 Vital Signs

Vital signs will be measured on Day 1 (M0), Day 30 (M1), Day 90 (M3), Day 120 (M4), and Day 270 (M9). These will include (but are not limited to) the measurement of systolic blood pressure/diastolic blood pressure, heart rate, and body temperature.

# 9.1.6 Immunogenicity Assessments

Blood samples for immunogenicity assessments will be collected from subjects in the immunogenicity subset randomly selected using IRT prior to administration of the first vaccination (TDV or placebo) (Day 1 [M0]), at 1 month (Day 120 [M4]) and at 6 months (Day 270 [M9]) after the second vaccination. Refer to Appendix D.

All samples will be collected in accordance with acceptable laboratory procedures. All blood samples will be processed and stored at the trial site as detailed in the Laboratory Guidelines.

# 9.1.7 Safety Assessments

Safety assessments will include collection and recording of solicited local (injection site) and systemic AEs, unsolicited AEs (non-serious AEs and SAEs), and MAAEs. Refer to Section 10.1 for safety definitions. Details on collection and reporting of AEs are in Section 10.5.

# 9.1.8 Contraception and Pregnancy Avoidance Procedure

For female subjects of childbearing potential, serum or urine pregnancy testing will be performed prior to vaccination at Day 1 (M0) and Day 90 (M3). Additional pregnancy tests may be performed during the trial if deemed necessary by the Investigator. Females of childbearing potential who are sexually active will be reminded during trial visits to adhere to acceptable contraceptive methods up to 6 weeks post second trial vaccination at Day 90 (M3). Subjects will be provided with information on acceptable methods of contraception as part of the subject informed consent process and will be asked to sign a consent form stating that they understand the requirements for avoidance of pregnancy and donation of ova. During the course of the trial, subjects of childbearing potential will receive continued guidance with respect to the avoidance of pregnancy as part of the trial procedures (Section 2.1); see also Section 7.2.

# 9.1.9 Pregnancy

To ensure subject safety and the safety of the unborn child, each pregnancy in a subject having received a trial vaccine must be reported to the Sponsor within 24 hours of the site learning of its occurrence. If the subject becomes pregnant during the trial, she will not receive any further doses of any Sponsor-supplied trial vaccine. The pregnancy must be followed to determine outcome, including spontaneous or voluntary termination, details of birth, and the presence or absence of

any birth defects, congenital abnormalities, or maternal and/or newborn complications. This follow-up should occur even if the intended duration of safety follow-up for the trial has ended.

Any pregnancy occurring following trial vaccine administration should be reported immediately, using a pregnancy notification form, to the safety contact listed in the Investigator Site File.

Should the pregnancy occur after administration of a blinded trial vaccine, the Investigator must inform the subject of their right to receive information regarding TDV or placebo assignment. If the subject chooses to receive unblinded information regarding TDV or placebo, the individual blind should be broken by the Investigator and procedures must be followed as described in Section 8.5.

# 9.1.10 Documentation of Subjects who are not Randomized

Investigators must account for all subjects who sign an informed consent form. If the subject is found to be not eligible at this visit, the Investigator should complete the eCRF. The IRT supplier should be contacted as a notification of non-randomization.

The primary reason for non-randomization is recorded in the eCRF using the following categories:

- Screen failure (did not meet one or more inclusion criteria or did meet one or more exclusion criteria).
- Withdrawal by subject.
- Trial terminated by Sponsor.
- Other (specify reason).

Subject numbers assigned to subjects who fail screening should not be reused.

# 9.2 Monitoring Subject Compliance to TDV or Placebo Administration

The Investigator or Investigator's designee records all injections of trial vaccine given to the subject in the eCRF.

# 9.3 Schedule of Observations and Procedures

The schedule for all trial-related procedures for all evaluations is shown in Section 2.1. Assessments should be completed at the designated visit/time point(s).

# 9.3.1 Pre-Vaccination Procedures (Day 1 [M0] and Day 90 [M3])

- Before performing any trial procedure, the signed informed consent form needs to be obtained. Refer to Section 9.1.1.
- 2. Check inclusion and exclusion criteria. Refer to Sections 7.1 and 7.2.
- 3. Collect demographic data. Refer to Section 9.1.2.

- 4. Collect medical history, prior medications/vaccinations, and concomitant medications. Refer to Section 9.1.2.
- 5. Review of systems: Review of systems is a structured interview that questions the subject regarding any complaints they have experienced across each organ system.
- 6. Perform a complete physical examination. Refer to Section 9.1.4.
- 7. Check vital signs. Refer to Section 9.1.5
- 8. Perform pregnancy testing (serum or urine) for female subjects of child bearing age. Refer to Section 9.1.9.
- 9. Provide female subjects of child bearing age with information on acceptable methods of contraception. Refer to Section 9.1.8.
- 10. Randomize the subject (Day 1 [M0]). Refer to Section 9.1.3.
- 11. Collect a pre-vaccination blood sample (Day 1 [M0]) from subjects included in the immunogenicity subset. Refer to Section 9.1.6.

Blood should be taken from the subject using an aseptic venipuncture technique for serological immunogenicity testing. Refer to the detailed collection and handling procedures outlined in the Procedures Manuals.

# 9.3.2 Vaccination Procedures (Day 1 [M0] and Day 90 [M3])

- 1. Confirm eligibility of the subject (Day J [M0]); see Section 7.1 and Section 7.2, or confirm that the subject does not meet any criteria for delaying or cancelling additional trial vaccination (Day 90 [M3]); see Section 7.3.
- 2. Administer the vaccine. Refer to Section 8.1.3.
- 3. Note: Trial vaccines (ie, TDV and placebo) will be dispensed by using IRT (see Section 8.2); packaging of the trial vaccines will be identical (see Section 8.1.1).

# 9.3.3 Post Vaccination Procedures (Day 1 [M0] and Day 90 [M3])

1. Careful training of the subject on how to measure local AEs and body temperature, how to complete the diary card and how often to complete the diary card. Training should be directed at the individual(s) who will perform the measurements of local AEs and those who will enter the information into the diary card. This individual may or may not be the subject, but if a person other than the subject enters information into the diary card, this person's identity must be documented in the trial file and this person must receive training on the diary card. Training of the subject on how to measure an injection site AE should be performed while the subject is under observation after vaccination.

# Diary card instructions must include the following:

• The subject must understand that timely completion of the diary card on a daily basis is a critical component of trial participation. The subject should also be instructed to write clearly and to complete the diary card in pen. Any corrections to the diary card that are performed by the person completing the diary card should include a single strikethrough line with a brief explanation for any change and be initialed and dated.

#### Please note:

- Diary cards will be the only source document allowed for remote collection of solicited local and systemic AEs (including body temperature measurements). The following additional rules apply to the documentation of safety information collected by diary card:
- The diary card should be reviewed with the subject.
- No corrections or additions to the diary card will be allowed after it is reviewed with the Investigator/designee.
- Any data that are identified as implausible or incorrect, and confirmed by the subject to be a transcription error should be corrected by the subject or the subject's legally acceptable representative on the diary card (the correction should include a single strikethrough line and should be initialed and dated by the subject).
- Any blank or illegible fields on the diary card not otherwise corrected as above will be missing in the eCRF.
- Relevant site personnel must enter all readable entries on the diary card into the eCRF.
- Any newly described solicited safety information should be added to the diary card by the subject and initialed and dated. Any new unsolicited safety information would be recorded in the subject source document as a verbally reported event and therefore captured as an AE and recorded in the Adverse Event eCRF.
- Starting on the day of vaccination, the subject will check for specific types of events at the injection site (solicited local AEs), any specific generalized symptoms (solicited systemic AEs), body temperature (any method), any other symptoms or change in the subject's health status, and any medications taken (excluding vitamins and minerals). These solicited AEs and body temperature will be recorded in the diary. Assessments should preferably take place in the evening at day's end.
- Body temperature measurement is to be performed using the thermometer provided by the site. If the subject feels unusually hot or cold during the day, the subject should check their temperature. If the subject has a fever, the highest body temperature observed that day should be recorded on the diary card.
- The measurement of solicited local AEs (erythema, swelling, and induration) is to be performed using the ruler provided by the site.

- The collection on the diary card of solicited local (injection site) AEs and solicited systemic AEs (including body temperature) will continue for a total of 7 days and 14 days, respectively, following each trial vaccination. Persistent/prolonged solicited local or systemic AEs continuing on Day 8 and Day 15 respectively, following each trial vaccination will be recorded in the subject source document as a verbally reported event and therefore captured as an AE and recorded in the Adverse Event eCRF. Refer to Section 10.4.2.
- 2. Provide female subjects of childbearing age with information on acceptable methods of contraception. Refer to Section 9.1.8.
- 3. Collect and record unsolicited AEs. Refer to Section 10.4.1.
- 4. Collect and record MAAEs. Refer to Section 10.4.3.
- 5. Collect and record SAEs. Refer to Section 10.4.4

After each trial vaccination, the subject will be observed for at least 30 minutes including observation for unsolicited AEs (non-serious and serious), solicited AEs, and body temperature measurement. Information should be recorded in the electronic data capture (EDC) system. The Investigator or delegate will take the opportunity to remind the subject how to measure solicited AEs and body temperature as part of this observation period. All safety data will be collected in the subject's source documents.

6. The site should schedule the next trial activity with the subject.

The subject will receive a written reminder of the next planned trial activity. The subject will be reminded to complete the diary card daily and to contact the site if there are any questions and to contact the site immediately (or as soon as the subject is medically stable) if the subject has a medical condition that leads to a hospitalization or an emergency room visit or is otherwise perceived as serious. All contact details will be provided to the subject.

# 9.3.4 Clinic Visits after Vaccination (Day 30 [M1], Day 120 [M4], and Day 270 [M9])

Clinic visits that do not include a vaccination will be performed on Day 30 (M1), Day 120 (M4), and Day 270 (M9). These visits should occur at least 29 Days after the first and second vaccination on Day 1 (M0) and Day 90 (M3).

- 1. Interview the subject and check the diary card (Day 30 [M1], and Day 120 [M4]). Refer to Section 9.3.3.
- 2. Perform a targeted physical examination. Refer to Sections 9.1.4 and 9.1.5.
- 3. Check vital signs. Refer to Section 9.1.5.
- 4. Provide pregnancy avoidance guidance to females of childbearing potential. Refer to Section 9.1.8.
- 5. Provide female subjects of childbearing age with information on acceptable methods of contraception. Refer to Section 9.1.8.

- 6. Record persistent/prolonged solicited AEs (Day 30 [M1], and Day 120 [M4]). Refer to Sections 9.3.3 and 10.4.2.
- 7. Record unsolicited AEs (Day 30 [M1], and Day 120 [M4]). Refer to Section 10.4.1.
- 8. Record and collect MAAEs and SAEs. Refer to Sections 10.4.3 and 10.4.4.
- 9. Collect a blood sample from subjects included in the immunogenicity subset (Day 120 [M4], and Day 270 [M9]). Refer to Section 9.1.6.

Blood should be taken from the subject using an aseptic venipuncture technique for serological immunogenicity testing. Refer to the detailed collection and handling procedures outlined in the Procedures Manuals.

10. The site should schedule the next trial activity clinic visit with the subject.

The subject will receive a written reminder of the next planned trial activity. The subject will be reminded to contact the site if there are any questions and to contact the site immediately (or as soon as the subject is medically stable) if the subject has a medical condition that leads to a hospitalization or an emergency room visit.

# 9.3.5 Final (End of Trial) Visit

The Final Visit will be performed on Day 270 (M9). If a subject terminates earlier, end of trial visit procedures should be performed if possible. For all subjects receiving trial vaccine (ie, TDV or placebo), the Investigator must complete the "End of Trial" eCRF page.

# 9.3.6 Post-Trial Care

No post-trial care will be provided.

# 9.4 Biological Sample Retention and Destruction

In this trial, specimens for immune response testing will be collected as described in Section 9.1.6. After blood draw and serum processing, the serum samples will be preserved and retained at a central laboratory contracted by the Sponsor for this purpose for up to but not longer than 20 years or as required by applicable law. The Sponsor has put into place a system to protect the subjects' personal information to ensure optimal confidentiality and defined standard processes for sample and data collection, storage, analysis, and destruction.

Serum samples will be used for the analyses defined in this protocol, but can also, with permission from the subject, be used to assess, improve or develop tests related to dengue or other disease(s) or the vaccine(s) under trial that will allow more reliable measurement of the response to the vaccine(s).

#### 10.0 ADVERSE EVENTS

#### 10.1 Definitions

#### 10.1.1 Adverse Events

An AE is defined as any untoward medical occurrence in a clinical investigation subject administered a trial vaccine; it does not necessarily have to have a causal relationship with trial vaccine administration.

An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the administration of a trial vaccine whether or not it is considered related to the trial vaccine.

AEs will be graded by the Investigator in the following manner:

| Mild | Grade 1 | • | Awareness of symptoms that are easily tolerated, causing minimal discomfort and not interfering with everyday activities. Relieved with or without symptomatic treatment. |
|---|---|---|---|
| Moderate | Grade 2 | • | Sufficient discomfort is present to cause interference with normal activity. Only partially relieved with symptomatic treatment. |
| Severe | Grade 3 | • | Extreme distress, causing significant impairment of functioning or incapacitation. Prevents normal everyday activities. Not relieved with symptomatic treatment |

# **10.1.2** Solicited Adverse Events

The occurrence of selected indicators of safety will be measured/collected for 7 days (solicited local [injection site] AEs) and 14 days (solicited systemic AEs) following administration of each trial vaccine dose (including the day of administration) and will be recorded on the "Local and Systemic Reactions" eCRF page as applicable and as listed in Table 10.a. These will be summarized in the final report under the category "solicited AEs" to differentiate them from other AEs which were not solicited. Any solicited local or systemic AE observed as continuing on Day 8 and Day 15, respectively, following each trial vaccination will be recorded as an AE on the Adverse Event eCRF for follow-up. For these persistent/prolonged solicited AEs the end date will be captured on the Adverse Event eCRF to permit a separate analysis from the unsolicited AEs (see Section 10.4.2).

Table 10.a Local and Systemic AEs

| Local AEs (injection site): | Pain | |
|-------------------------------------------------|-----------|------|
| | Erythema | |
| | Swelling | |
| Systemic AEs (adult/adolescent/child ≥6 years): | Fever (a) | 70. |
| | Headache | |
| | Asthenia | |
| | Malaise | CO. |
| | Myalgia | |
| | | 4 1. |

<sup>(</sup>a) Fever is defined as body temperature greater than or equal to 38°C (100.4°F) regardless of method used [17].

The intensity of solicited safety parameters will be assessed as described in Table 10.b.

**Table 10.b** Solicited Safety Parameters

| Tuble 10.5 Soller | tea Salety 1 alai | neter 5 |
|---|---|---|
| Adverse Event | Intensity grade | Severity/Intensity |
| Pain at injection site | 0 | None |
| | 1 | Mild: No interference with daily activity |
| | 2 | Moderate: Interference with daily activity with or without treatment |
| | 3 | Severe: Prevents daily activity with or without treatment |
| Erythema at injection | 0 | <25 mm |
| site (a) | 1 | Mild: ≥25 – ≤50 mm |
| | 2 | Moderate: $>$ 50 – $\leq$ 100 mm |
| | 3 | Severe:>100 mm |
| Swelling at injection | 0 | <25 mm |
| site (a) | 1 | Mild: $\geq 25 - \leq 50 \text{ mm}$ |
| | 2 | Moderate: >50 – ≤100 mm |
| | 3 | Severe: >100 mm |
| Headache | 0 | None |
| | 1 | Mild: No interference with daily activity |
| | $\sim$ 2 | Moderate: Interference with daily activity with or without treatment |
| | 3 | Severe: Prevents normal activity with or without treatment |
| Asthenia | 0 | None |
| | 1 | Mild: No interference with daily activity |
| 1.0 | 2 | Moderate: Interference with daily activity |
| | 3 | Severe: Prevents daily activity |
| Malaise \(\sigma^*\) | 0 | None |
| CO. | 1 | Mild: No interference with daily activity |
| Ho | 2 | Moderate: Interference with daily activity |
| Υ',0, | 3 | Severe: Prevents daily activity |
| Myalgia | 0 | None |
| 0 | 1 | Mild: No interference with daily activity |
| } | 2 | Moderate: Interference with daily activity |
| | 3 | Severe: Prevents daily activity |
| Fever (b) | Record body tempe | · · · |
| / \ ~ | | |

<sup>(</sup>a) Subjects are to record greatest surface diameter in mm on the diary card.

<sup>(</sup>b) Fever is defined as greater than or equal to 38°C (100.4°F) regardless of method used [17].

# 10.1.3 Medically Attended Adverse Events

MAAEs are defined as AEs leading to an unscheduled visit to or by a healthcare professional including visits to an emergency department, but not fulfilling seriousness criteria.

#### **10.1.4 Serious Adverse Events**

An SAE is defined as any untoward medical occurrence that:

- 1. Results in DEATH.
- 2. Is LIFE THREATENING.
- The term "life threatening" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.
- 3. Requires inpatient HOSPITALIZATION or prolongation of existing hospitalization.
- 4. Results in persistent or significant DISABILITY/INCAPACITY.
- 5. Leads to a CONGENITAL ANOMALY/BIRTH DEFECT in the offspring of a subject.
- 6. Is an IMPORTANT MEDICAL EVENT that satisfies any of the following:
- May require intervention to prevent items 1 through 5 above.
- May expose the subject to danger, even though the event is not immediately life threatening or fatal or does not result in hospitalization.

# 10.2 Causality of Adverse Events

Relatedness (causality) to vaccine will also be assessed by the Investigator. The relationship of each AE, including solicited systemic AEs (solicited local AEs are considered as related) to trial vaccine(s) will be assessed using the following categories:

| Related: | There is suspicion that there is a relationship between the trial vaccine and the AE |
|---|---|
| | (without determining the extent of probability); there is a reasonable possibility that the |
| | trial vaccine contributed to the AE. |
| Not Related: | There is no suspicion that there is a relationship between the trial vaccine and the AE; |
| 7,0 | there are other more likely causes and administration of the trial vaccine is not suspected |
| Tec | to have contributed to the AE. |

# 10.2.1 Relationship to Trial Procedures

Relationship (causality) to trial procedures should be determined for all AEs.

The relationship should be assessed as "Yes" if the Investigator considers that there is reasonable possibility that an event is due to a trial procedure. Otherwise, the relationship should be assessed as "No".

#### Outcome of Adverse Events

| Resolved: | The subject has fully recovered from the event or the condition has returned to the level observed at Baseline. |
|---|---|
| Resolving: | The event is improving but the subject is still not fully recovered. |
| Not resolved: | The event is ongoing at the time of reporting and the subject has still not recovered. |
| Resolved with sequelae: | As a result of the AE, the subject suffered persistent and significant disability/incapacity (eg, became blind, deaf or paralysed). |
| Fatal: | The subject died due to the event. If the subject died due to other circumstances than the event, the outcome of the event per se should be stated otherwise (eg, Not Resolved or Resolving). |
| Unknown: | If outcome is not known or not reported. |

# 10.3 Additional Points to Consider for Adverse Events

An untoward occurrence generally may:

- Indicate a new diagnosis or unexpected worsening of a pre-existing condition. Intermittent events for pre-existing conditions or underlying disease should not be considered as AEs.
- Necessitate therapeutic intervention.
- Require an invasive diagnostic procedure.
- Require vaccine discontinuation or a change in concomitant medication.
- Be considered unfavorable by the Investigator for any reason.

Diagnoses vs. signs and symptoms:

• Each event should be recorded to represent a single diagnosis. Accompanying signs (including abnormal laboratory values) or symptoms should NOT be recorded as additional AEs. If a diagnosis is unknown, signs or symptoms should be recorded appropriately as AEs.

# Worsening of AEs:

- If the subject experiences a worsening or complication of an AE after starting administration of the trial vaccine, the worsening or complication should be recorded as a new AE. Investigators should ensure that the AE term recorded captures the change in the condition (eg, "worsening of...").
- If the subject experiences a worsening or complication of an AE after any change in trial vaccine, the worsening or complication should be recorded as a new AE. Investigators should ensure that the AE term recorded captures the change in the condition (eg, "worsening of...").

# Changes in severity of AEs:

• If the subject experiences changes in severity of an AE, the event should be captured once with the maximum severity recorded.

# Preplanned surgeries or procedures:

 Preplanned procedures (surgeries or therapies) that were scheduled prior to signing of informed consent form are not considered AEs. Complications resulting from any planned surgery should be reported as AEs.

# Elective surgeries or procedures:

• Elective procedures performed where there is no change in the subject's medical condition should not be recorded as AEs, but should be documented in the subject's source documents. Complications resulting from an elective surgery should be reported as AEs.

#### 10.4 Procedures

# 10.4.1 Collection and Reporting of Adverse Events

All AEs, whether considered related to the use of the trial vaccine or not, must be monitored until symptoms subside and any abnormal laboratory values have returned to Baseline, or until there is a satisfactory explanation for the changes observed, or until death, in which case a full pathologist's report should be supplied, if possible. All findings must be reported on an Adverse Event eCRF and on the SAE form, if necessary (see Section 10.4.2). All findings in subjects experiencing AEs must also be reported in the subject's source documents. Any unsolicited AEs will be collected for 28 days (day of vaccination + 27 days) following each TDV/placebo dose during site visits via interview; AEs leading to withdrawal or discontinuation will be collected throughout the trial.

The following information will be documented for each event:

- Reported term for the AE.
- Start and end date.
- Serious (Y/N).
- Severity,
- Investigator's opinion of the causality (relationship) between the event and administration of trial vaccine(s) ("related" or "not related").
- Investigator's opinion of the causality (relationship) to trial procedure(s), including the details of the suspected procedure.
- Action taken with the trial vaccine.
- Outcome of event.

# 10.4.2 Collection and Reporting of Solicited Adverse Events

The occurrence of selected indicators of safety will be collected on diary cards by the subjects for 7 days (solicited local [injection site] AEs) and 14 days (solicited systemic AEs) following administration of each trial vaccine dose (including the day of administration) and will be recorded on the "Local and Systemic AEs" eCRF, as applicable. These will be summarized in the final report under the category "solicited adverse events" to differentiate them from unsolicited AEs. Any solicited local (injection site) or systemic AE observed as continuing on Day 8 and Day 15, respectively, following each trial vaccination will be additionally recorded as an AE on the Adverse Event eCRF for follow-up. For these persistent/prolonged solicited AEs the end date will be captured on the Adverse Event eCRF to permit a separate analysis from the unsolicited AEs. Any solicited local (injection site) or systemic AE that resolves before 8 days and 15 days, respectively, following each trial dose administration, but that recurs at a later time (ie, if discontinues), will be recorded as an unsolicited AE on the Adverse Event eCRF.

Any solicited AE that meets any of the following criteria must be entered as an AE on the Adverse Event eCRF.

- Solicited local or systemic AEs that lead the subject to withdraw from the trial.
- Solicited local or systemic AEs that lead to the subject being withdrawn from the trial by the Investigator.
- Solicited local and systemic AEs that otherwise meet the definition of an SAE (see Section 10.1.2).

# 10.4.3 Collection and Reporting of Medically Attended Adverse Events

MAAEs will be collected for the trial duration: occurring from the first vaccination at Day 1 (M0) up to 6 months post second dose at Day 90 (M3), and will be collected by interview at Day 30 (M1), Day 90 (M3), Day 120 (M4), and Day 270 (M9) and must be recorded as an AE on the Adverse Event eCRF.

# 10.4.4 Collection and Reporting of Serious Adverse Events

Collection of SAEs will commence from the time that the subject first receives the trial vaccine (Day 1 [M0]). Routine collection of SAEs will continue until the end of the trial (Day 270 [M9]).

SAEs should be reported according to the following procedure:

A Sponsor SAE form must be completed, in English, and signed by the Investigator immediately or within 24 hours of first onset or notification of the event. The information should be completed as fully as possible but contain, at a minimum:

- A short description of the event and the reason why the event is categorized as serious.
- Subject identification number.
- Investigator's name.

The SAE form should be transmitted within 24 hours to the attention of the contact(s) in the list provided to each site.

10.5 Follow-up Procedures

#### 10.5.1 Adverse Events

All AEs will be monitored until resolution or a stable status is reached or until a formal diagnosis can be made or until the end of the trial, whichever occurs first. This could potentially be followed outside of this trial or in a planned extension trial.

#### **10.5.2** Serious Adverse Events

If information not available at the time of the first report becomes available at a later date, the Investigator should complete a follow-up SAE form or provide other written documentation and fax it immediately within 24 hours of receipt. Copies of any relevant data from the hospital notes (eg, laboratory tests, discharge summary, postmortem results) should be sent to the Sponsor.

All SAEs should be followed up until resolution or permanent outcome of the event or is otherwise explained. The timelines and procedure for follow-up reports are the same as those for the initial report.

# 10.5.3 Safety Reporting to Investigators, Institutional Review Boards, and Regulatory **Authorities**

The Sponsor or designee will be responsible for the reporting of all Suspected Unexpected Serious Adverse Reactions (SUSARs) and any other applicable SAEs to regulatory authorities, Investigators and IRBs, as applicable, in accordance with national regulations in the countries where the trial is conducted. Relative to the first awareness of the event by/or further provision to the Sponsor's designee, SUSARs will be submitted within 7 days for fatal and life-threatening events and 15 days for other SUSARs, unless otherwise required by national regulations. The Sponsor will also prepare an expedited report for other safety issues where these might materially alter the current benefit-risk assessment of an investigational medicinal product or that would be sufficient to consider changes in the trial vaccine administration or in the overall conduct of the trial. The investigational site also will forward a copy of all expedited reports to their IRB in accordance with national regulations.

# 10.5.4 Post-Trial Events

Any SAE that occurs outside of the protocol-specified observation period or after the end of the trial but considered to be caused by the trial vaccine(s) must be reported to the Sponsor. These SAEs will be processed by the Sponsor's Pharmacovigilance Department. Instructions for how to submit these SAEs will be provided in a handout in the Investigator Site File.

#### TRIAL-SPECIFIC REQUIREMENT(S) 11.0

#### 11.1 **Trial-Specific Committees**

# 11.1.1 Data Monitoring Committee

relins of Use ogr Properly of Takeda. For noncommercial use only and subject to the application of takeda. A DMC will have oversight of this clinical trial. The DMC functions at a Takeda dengue program

## 12.0 DATA HANDLING AND RECORDKEEPING

The full details of procedures for data handling will be documented in the Data Management Plan. AEs, medical history, and concurrent conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA, System Organ Class [SOC], High Level Group Term, High Level Term, Low Level Term, Preferred Term [PT], and their corresponding descriptive terms). Drugs will be coded using the WHO Drug Dictionary.

## 12.1 Electronic CRFs (eCRF)

Completed eCRFs are required for each subject who provides a signed informed consent.

The Sponsor or designee will supply investigative sites with access to eCRFs. The Sponsor will make arrangements to train appropriate site staff in the use of the eCRF. eCRFs must be completed in English.

After completion of the entry process, computer logic checks will be run to identify items, such as inconsistent dates, missing data, and questionable values. Queries may be issued by Sponsor personnel (or designees) and will be answered by the site.

Corrections to eCRFs are recorded in an audit trail that captures the old information, the new information, identification of the person making the correction, the date the correction was made, and the reason for change.

The Principal Investigator or designee must review the eCRFs for completeness and accuracy and must sign and date the appropriate eCRFs as indicated. Furthermore, the Investigator must retain full responsibility for the accuracy and authenticity of all data entered on the eCRFs.

eCRFs will be reviewed for completeness and acceptability at the trial site during periodic visits by trial monitors. The Sponsor or designee will be permitted to review the subject's medical and hospital records pertinent to the trial to ensure accuracy of the eCRFs. The completed eCRFs are the sole property of the Sponsor and should not be made available in any form to third parties, except for authorized representatives of appropriate governmental health or regulatory authorities, without written permission of the Sponsor.

# 12.2 Record Retention

The Investigator agrees to keep the records stipulated in Section 12.0 and those documents that include (but are not limited to) the trial-specific documents, the identification log of all participating subjects, medical records. Temporary media such as thermal sensitive paper should be copied and certified, source worksheets, all original signed and dated informed consent forms, subject authorization forms regarding the use of personal health information (if separate from the informed consent or forms), electronic copy of eCRFs, including the audit trail, and detailed records of vaccine disposition to enable evaluations or audits from regulatory authorities, the Sponsor or designees. Furthermore, ICH E6 Section 4.9.5 requires the Investigator to retain essential documents specified in ICH E6 (Section 8) until at least 2 years after the last approval of a marketing application for a specified vaccine indication being investigated or, if an application is

not approved, until at least 2 years after the investigation is discontinued and regulatory authorities are notified. In addition, ICH E6 Section 4.9.5 states that the trial records should be retained until an amount of time specified by applicable regulatory requirements or for a time specified in the Clinical Trial Site Agreement between the Investigator and Sponsor.

ord rete, ore disposition and antique applications and allowed the property of takeda. For non-commercial use only and allowed the property of takeda. For non-commercial use only and allowed the property of takeda. Refer to the Clinical Trial Site Agreement for the Sponsor's requirements on record retention. The Investigator should contact and receive written approval from the Sponsor before disposing of any

## 13.0 STATISTICAL METHODS

## 13.1 Statistical and Analytical Plans

A statistical analysis plan (SAP) will be prepared and finalized prior to the database lock and unblinding of subject's trial vaccine assignment. This document will provide further details regarding the definition of analysis variables and analysis methodology to address all trial objectives.

A blinded review of data will be conducted prior to unblinding of subject's trial vaccine assignment. This review will assess the accuracy and completeness of the trial database, subject evaluability, and appropriateness of the planned statistical methods.

# 13.1.1 Analysis Sets

Safety set: The safety set will consist of all subjects who received at least 1 dose of trial vaccine.

**Full analysis set (FAS):** The FAS will include all randomized subjects in the immunogenicity subset who received at least 1 dose of trial vaccine and for whom a valid pre-dose and at least one valid post-dose blood sample is taken.

**Per–protocol set (PPS):** The PPS will exclude all subjects seropositive for dengue virus at Baseline and will include all subjects in the FAS who have no major protocol violations. The major protocol violation criteria will be defined as part of the blinded data review prior to the unblinding of the trial vaccine assignment. The categories of major protocol violations include: (1) not meeting selected entry criteria, (2) not receiving a the correct randomly assigned trial vaccine or placebo, (3) receiving prohibited therapies, (4) not receiving 2 doses of trial vaccine or receiving the second trial dose inadmissibly outside of the visit window, and (5) other major protocol violations that may be identified during blinded data reviews.

All summaries and analyses of safety data will be based on subjects in the safety set. The primary immunogenicity analyses will be based on the PPS; additional immunogenicity analyses may be provided based on the FAS.

# 13.1.2 Analysis of Demographics and Other Baseline Characteristics

Age, gender, race, and other Baseline characteristics will be summarized descriptively by trial group for all randomized subjects.

# 13.1.3 Immunogenicity Analysis

An immunogenicity subset of 616 subjects (TDV groups: 176 subjects each and placebo group: 88 subjects) will be randomly selected for the immunogenicity analyses (ie, the immunogenicity subset).

For the primary and secondary immunogenicity endpoints (ie, GMTs of neutralizing antibodies and seropositivity rates for each of the 4 dengue serotypes), descriptive statistics and 95% CIs will

be provided by trial group for each applicable visit (Day 120 [M4] and Day 270 [M9]). Seropositivity is defined as a reciprocal neutralizing titer ≥10.

The primary endpoint will evaluate lot-to-lot consistency at Day 120 (M4). For each serotype, an analysis of variance (ANOVA) model on the natural logarithms of titers of dengue neutralizing antibodies will include data from subjects in Groups 1-3 with trial group as a factor. A 95% CI will be provided for the 3 pairwise comparisons of log-transformed GMTs. The CIs will be back-transformed in order to report 95% CIs of the ratios in the original scale. For each pairwise comparison, equivalence of immune responses will be established if the 95% CI for the ratio is contained between equivalence margins of 0.5 and 2.0. Lot-to-lot consistency will be concluded if equivalence of immune responses is established for all pairwise comparisons and all 4 dengue serotypes. For the secondary endpoint of GMT at Day 270 (M9), a similar model will be fit.

For the secondary endpoint of seropositivity, 95% CIs for the difference in proportions between groups of interest for each dengue serotype at each applicable visit will be constructed using the Newcombe and Wilson method.

The primary immunogenicity analyses will be based on the PPS; other immunogenicity analyses may be provided based on the FAS.

# 13.1.4 Safety Analysis

All safety data will be summarized by trial group using the safety set.

## Solicited AEs

In all subjects, the presence and severity (Grade) of solicited local AEs (injection site pain, injection site erythema and injection site swelling) and solicited systemic AEs (fever, asthenia, malaise, headache and myalgia) will be collected for 7 days and 14 days, respectively, following each vaccination (including the day of vaccination) via collection of diary cards.

For each solicited AE, the number and percentage of subjects with local AEs (injection site) and systemic AEs will be summarized by trial group and event severity for each day after each vaccination (ie, Day 1 through Day 7 for local AEs [injection site] AEs and Day 1 through Day 14 for systemic AEs), and overall. Summaries of first onset of each event and the number of days subjects reported experiencing each event will also be provided. For subjects with more than 1 episode of the same event, the maximum severity will be used for tabulations.

Persistent/prolonged solicited local or systemic AEs continuing on Day 8 and Day 15, respectively, following each trial vaccination will be assessed separately. Unless otherwise specified these AEs will not be included in the analyses/tabulations of unsolicited AEs and will have separate listings.

## Unsolicited AEs

Unsolicited AEs will be assessed for 28 days following each TDV/placebo dose (day of vaccination + 27 days).

In all subjects, unsolicited AEs will be coded using the MedDRA and summarized by SOC and PT for each trial group. AEs leading to trial or vaccine withdrawal will also be summarized for the duration of the trial.

Unsolicited AEs will be summarized as follows: by PT including events with frequency greater than a pre-defined frequency (the percentage will be specified in the SAP); by SOC and PT; by SOC, PT, and severity; and by SOC, PT, and relationship to the investigational vaccine. Subjects reporting more than 1 occurrence for the term (level) being summarized will be counted only once.

# **MAAEs**

In all subjects, MAAEs will be collected throughout the trial. MAAEs will be coded using MedDRA and summarized by SOC and PT for each trial group.

# **SAEs**

In all subjects, SAEs will be collected throughout the trial. SAEs will be coded using MedDRA, and summarized by SOC and PT for each trial group.

# 13.2 Interim Analysis and Criteria for Early Termination

No interim analyses are planned.

# 13.3 Determination of Sample Size

It is assumed that the natural logarithms of titers of neutralizing antibodies for each of the 4 dengue serotypes are distributed as independent normal distributions, with standard deviations of 1.35, 0.86, 1.21, and 1.27, respectively. A sample size of 137 evaluable subjects in each of the 3 TDV groups (ie, Groups 1-3) is sufficient to achieve approximately 90% overall power for establishing lot-to-lot consistency in terms of equivalence of immune responses to 3 consecutive TDV lots based on the 95% CIs of the titer ratios, using equivalence margins of 0.5 and 2.0. This sample size assumes no variation among the 3 TDV lots; that is, for each serotype, the true ratio of GMT is 1.0 between the first and second lots and between the second and third lots.

Further adjusted for approximately 20% dropouts and non-evaluable subjects, the required sample size to evaluate lot-to-lot consistency is approximately 176 subjects for each TDV group and 88 subject for the placebo group, given 2:2:2:1 randomization ratio between trial groups and taking into account ratio between the immunogenicity subset and its complement. Therefore, the immunogenicity subset will include 616 subjects.

To ensure sufficient size of the safety database in the dengue non-endemic regions, overall sample size for the trial is 924 subjects: 264 for each TDV group and 132 for the placebo group.

# 14.0 QUALITY CONTROL AND QUALITY ASSURANCE

# **14.1** Trial-Site Monitoring Visits

Monitoring visits to the trial site will be made periodically during the trial to ensure that all aspects of the protocol are followed. Source documents will be reviewed for verification of data recorded on the eCRFs. Source documents are defined as original documents, data, and records. The Investigator and institution guarantee access to source documents by the Sponsor or designee (contract research organization) and by the IRB.

All aspects of the trial and its documentation will be subject to review by the Sponsor or designee (as long as blinding is not jeopardized), including but not limited to the Investigator's Binder, trial vaccine, subject medical records, informed consent form documentation, documentation of subject authorization to use personal health information (if separate from the informed consent forms), and review of eCRFs and associated source documents. It is important that the Investigator and other trial personnel are available during the monitoring visits and that sufficient time is devoted to the process.

### 14.2 Protocol Deviations

The Investigator should not deviate from the protocol, except where necessary to eliminate an immediate hazard to trial subjects. Should other unexpected circumstances arise that will require deviation from protocol-specified procedures, the Investigator should consult with the medical monitor (and IRB, as required) to determine the appropriate course of action. There will be no exemptions (a prospective approved deviation) from the inclusion or exclusion criteria.

# 14.3 Quality Assurance Audits and Regulatory Agency Inspections

The trial site also may be subject to quality assurance audits by the Sponsor or designees. In this circumstance, the Sponsor-designated auditor will contact the site in advance to arrange an auditing visit. The auditor may ask to visit the facilities where laboratory samples are collected, where the vaccine is stored and prepared, and any other facility used during the trial. In addition, there is the possibility that this trial may be inspected by regulatory agencies, including those of foreign governments (eg, the Food and Drug Administration [FDA], the United Kingdom Medicines and Healthcare Products Regulatory Agency, the Pharmaceuticals and Medical Devices Agency of Japan). If the trial site is contacted for an inspection by a regulatory body, the Sponsor should be notified immediately. The Investigator and institution guarantee access for quality assurance auditors to all trial documents as described in Section 14.1.

#### 15.0 ETHICAL ASPECTS OF THE TRIAL

SONJEE This trial will be conducted with the highest respect for the individual participants (ie, subjects) according to the protocol, the ethical principles that have their origin in the Declaration of Helsinki, and the ICH Harmonized Tripartite Guideline for GCP. Each Investigator will conduct the trial according to applicable local or regional regulatory requirements and align his or her conduct in accordance with the "Responsibilities of the Investigator" that are listed in Appendix A. The principles of Helsinki are addressed through the protocol and through appendices containing requirements for informed consent and Investigator responsibilities.

#### 15.1 **Institutional Review Board**

IRBs must be constituted according to the applicable local requirements of each participating region. The Sponsor or designee will require documentation noting all names and titles of members who make up the respective IRB If any member of the IRB has direct participation in this trial, written notification regarding his or her abstinence from voting must also be obtained. Those US sites unwilling to provide names and titles of all members due to privacy and conflict of interest concerns should instead provide a Federal Wide Assurance Number or comparable number assigned by the Department of Health and Human Services.

The Sponsor or designee will supply relevant documents for submission to the respective IRB for the protocol's review and approval. This protocol, the Investigator's Brochure, a copy of the informed consent form, and, if applicable, subject recruitment materials and/or advertisements and other documents required by all applicable laws and regulations, must be submitted to a central or local IRB for approval. The IRB's written approval of the protocol and subject informed consent form must be obtained and submitted to the Sponsor or designee before commencement of the trial (ie, before shipment of the Sponsor-supplied vaccine or trial specific screening activity). The IRB approval must refer to the trial by exact protocol title, number, and version date; identify versions of other documents (eg, informed consent form) reviewed; and state the approval date. The Sponsor will notify the site once the Sponsor has confirmed the adequacy of site regulatory documentation and, when applicable, the Sponsor has received permission from the competent authority to begin the trial. Until the site receives [notification] no protocol activities, including screening may occur.

Sites must adhere to all requirements stipulated by their respective IRB. This may include notification to the IRB regarding protocol amendments, updates to the informed consent form, recruitment materials intended for viewing by subjects, local safety reporting requirements, reports and updates regarding the ongoing review of the trial at intervals specified by the respective IRB, and submission of the Investigator's final status report to IRB. All IRB approvals and relevant documentation for these items must be provided to the Sponsor or designee.

Subject incentives should not exert undue influence for participation. Payments to subjects must be approved by the IRB and Sponsor.

#### 15.2 Subject Information, Informed Consent, and Subject Authorization

ns of Use Written consent documents will embody the elements of informed consent as described in the Declaration of Helsinki and the ICH Guidelines for GCP and will be in accordance with all applicable laws and regulations. The informed consent form, subject authorization form (if applicable), and subject information sheet (if applicable) describe the planned and permitted uses, transfers, and disclosures of the subject's personal and personal health information for purposes of conducting the trial. The informed consent form and the subject information sheet (if applicable) further explain the nature of the trial, its objectives, and potential risks and benefits, as well as the date informed consent is given. The informed consent form will detail the requirements of the participant and the fact that he or she is free/ to withdraw at any time without giving a reason and without prejudice to his or her further medical care.

The Investigator is responsible for the preparation, content, and IRB approval of the informed consent form and if applicable, the subject authorization form. The informed consent form, subject authorization form (if applicable), and subject information sheet (if applicable) must be approved by both the IRB and the Sponsor prior to use.

The informed consent form, subject authorization form (if applicable), and subject information sheet (if applicable) must be written in a language fully comprehensible to the prospective subject. It is the responsibility of the Investigator to explain the detailed elements of the informed consent form, subject authorization form (if applicable), and subject information sheet (if applicable) to the subject. Information should be given in both oral and written form whenever possible and in the manner deemed appropriate by the IRB.

The subject must be given ample opportunity to: (1) inquire about details of the trial and (2) decide whether or not to participate in the trial. If the subject determines he or she will participate in the trial, then the informed consent and subject authorization form (if applicable) must be signed and dated by the subject at the time of consent and prior to the subject entering into the trial. The subject should be instructed to sign using their legal names, not nicknames, using blue or black ballpoint ink. The Investigator must also sign and date the informed consent form and subject authorization (if applicable) at the time of consent and prior to subject entering into the trial; however, the Sponsor may allow a designee of the Investigator to sign to the extent permitted by applicable law.

Once signed, the original informed consent form, subject authorization form (if applicable), and subject information sheet (if applicable) will be stored in the Investigator's site file. The Investigator must document the date the subject signs the informed consent form in the subject's medical record and eCRF. Copies of the signed informed consent form, the signed subject authorization form (if applicable), and subject information sheet (if applicable) shall be given to the subject.

All revised informed consent forms must be reviewed and signed by the relevant subject in the same manner as the original informed consent form. The date the revised consent was obtained should be recorded in the subject's medical record and eCRF, and the subject should receive a copy of the revised informed consent form.

# 15.3 Subject Confidentiality

The Sponsor and designees affirm and uphold the principle of the subject's right to protection against invasion of privacy. Throughout this trial, a subject's source data will only be linked to the Sponsor's clinical trial database or documentation via a unique identification number. As permitted by all applicable laws and regulations, limited subject attributes, such as sex, age, or date of birth, and subject initials may be used to verify the subject and accuracy of the subject's unique identification number.

To comply with ICH Guidelines for GCP and to verify compliance with this protocol, the Sponsor requires the Investigator to permit its monitor or designee's monitor, representatives from any regulatory authority (eg, FDA, Medicines and Healthcare products Regulatory Agency, Pharmaceuticals and Medical Devices Agency), the Sponsor's designated auditors, and the appropriate IRBs to review the subject's original medical records (source data or documents), including, but not limited to, laboratory test result reports, electrocardiogram (ECG) reports, admission and discharge summaries for hospital admissions occurring during a subject's trial participation, and autopsy reports. Access to a subject's original medical records requires the specific authorization of the subject as part of the informed consent form process (see Section 15.2).

Copies of any subject source documents that are provided to the Sponsor must have certain personally identifiable information removed (ie. subject name, address, and other identifier fields not collected on the subject's eCRF).

# 15.4 Publication, Disclosure, and Clinical Trial Registration Policy

# 15.4.1 Publication and Disclosure

The results of this trial are expected to be published in a scientific journal. It is anticipated that clinical and laboratory co-Investigators will participate in authorship. The order of authorship and choice of journal will be proposed by the Sponsor to the Principal Investigators, to be eventually agreed upon by all authors. The data analysis center for this trial will provide the analyses needed for publication. Information regarding this trial will be posted on ClinicalTrials.gov.

# 15.4.2 Clinical Trial Registration

In order to ensure that information on clinical trials reaches the public in a timely manner and to comply with applicable law, regulation and guidance, the Sponsor will, at a minimum register all clinical trials conducted in subjects that it Sponsors anywhere in the world on ClinicalTrials.gov or other publicly accessible websites before trial initiation. The Sponsor contact information, along with Investigator's city, country, and recruiting status will be registered and available for public viewing.

## 15.4.3 Clinical Trial Results Disclosure

The Sponsor will post the results of this clinical trial, regardless of outcome, on ClinicalTrials.gov or other publicly accessible websites, as required by applicable laws and/or regulations.

Trial completion corresponds to the date on which the final subject was examined or received an intervention for the purposes of final collection of data for the primary outcome, whether the clinical trial concluded according to the pre-specified protocol or was terminated.

# 15.5 Insurance and Compensation for Injury

Each subject in the trial must be insured in accordance with the regulations applicable to the site where the subject is participating. If a local underwriter is required, then the Sponsor or Sponsor's Property of Takeda. For noncommercial use only and subject to the designee will obtain clinical trial insurance against the risk of injury to clinical trial subjects. Refer to the Clinical Trial Site Agreement regarding the Sponsor's policy on subject compensation and treatment for injury. If the Investigator has questions regarding this policy, he or she should

- Simmons CP, Farrar JJ, Nguyen v V, Wills B. Dengue. N Engl J Med. 2012;366(15):1423-32.
   Gubler DJ. Epidemic dengue/dengue hemorrhagic fever as a public health, social and economic problem in the 21st century. Trends Microbiol. 2002;10(2):100-3.
   Guzman MG, Kouri G. Dengue: an update. Lancet Infect Dis. 2002;2(1):22-42
   World Health C.
- 4. World Health Organization, 2018. Dengue and severe dengue. Fact Sheet. Available at: http://www.who.int/mediacentre/factsheets/fs117/en/ [Accessed 29 October 2018].
- 5. World Health Organization, 1997. Dengue hemorrhagic fever: diagnosis, treatment, prevention and control, 2nd Edition. Available at: http://www.who.int/csr/resources/publications/dengue/Denguepublication/en/ [Accessed 29 October 2018].
- 6. Dengue: Guidelines for Diagnosis, Treatment, Prevention And Control. Geneva: World Health Organization. 2009.
- 7. Halstead SB, Deen J. The future of dengue vaccines. Lancet. 2002;360(9341):1243-5.
- 8. Sanofi Pasteur, 2018. An informational website about dengue and dengue vaccination for media. Available at: http://www.dengue.info [Accessed 29 October 2018].
- 9. Hadinegoro SR, Arredondo-Garcia JL, Capeding MR, Deseda C, Chotpitayasunondh T, Dietze R, et al. Efficacy and Long-Term Safety of a Dengue Vaccine in Regions of Endemic Disease. N Engl J Med. 2015;373(13):1195-206.
- 10. Simmons CP. A Candidate Dengue Vaccine Walks a Tightrope. N Engl J Med. 2015;373(13):1263-4.
- 11. Yoksan S, Bhamarapravati N, Halstead S.B. Dengue virus vaccine development: study on biological markers of unclosed dengue 1-4 viruses serially passaged in primary kidney cells. In: TD St. George, BH Kay and J Blok (ed.), Arbovirus research in Australia. Proceedings of the 4th Symposium CSIRO/QIMR; 1986; Brisbane, Australia.
- 12. Huang CY, Butrapet S, Tsuchiya KR, Bhamarapravati N, Gubler DJ, and Kinney RM. Dengue 2 PDK-53 virus as a chimeric carrier for tetravalent dengue vaccine development. J Virol. 2003;77(21):11436-47.
- 13. Tetravalent Dengue Vaccine Candidate (TDV) Global Investigator's Brochure Edition 9, 20 July 2018.
- 14. Guidelines for independent lot release of vaccines by regulatory authorities. In: WHO Expert Committee on Biological Standardization. Sixty-first report. Geneva, World Health Organization, 2013 (WHO Technical Report Series, No. 978), Annex 2.
- 15. WHO Expert Committee on Biological Standardization. World Health Organization Tech Rep Ser 2013. 978:1-384.

- 16. World Health Organization. Reducing pain at the time of vaccination: WHO position paper—
- Kohl KS, Marcy SM, Blum M, Connell Jones M, Dagan R, Hansen J, et al. Fever after immunization: current concepts and improved future scientific understanding. Clin Infect Dis. 2004;39(3):389-94. after Clin Infeq and Subject to the addicable only and subject to the addicable only addicable only addicab 17. Kohl KS, Marcy SM, Blum M, Connell Jones M, Dagan R, Hansen J, et al. Fever after

## APPENDIX A RESPONSIBILITIES OF THE INVESTIGATOR

cable terms of Use Clinical research trials sponsored by the Sponsor are subject to ICH GCP and all the applicable local laws and regulations.

The Investigator agrees to assume the following responsibilities:

- 1. Conduct the trial in accordance with the protocol.
- 2. Personally conduct or supervise the staff who will assist in the protocol.
- 3. Ensure that trial related procedures, including trial specific (non-routine/non-standard panel) screening assessments are NOT performed on potential subjects, prior to the receipt of written approval from relevant governing bodies/authorities.
- 4. Ensure that all colleagues and employees assisting in the conduct of the trial are informed of these obligations.
- 5. Secure prior approval of the trial and any changes by an appropriate IRB that conform to 21 Code of Federal Regulations (CFR) Part 56, ICH, and local regulatory requirements.
- 6. Ensure that the IRB will be responsible for initial review, continuing review, and approval of the protocol. Promptly report to the IRB all changes in research activity and all anticipated risks to subjects. Make at least yearly reports on the progress of the trial to the IRB, and issue a final report within 3 months of trial completion.
- 7. Ensure that requirements for informed consent, as outlined in 21 CFR Part 50, ICH and local regulations, are met.
- 8. Obtain valid informed consent from each subject who participates in the trial, and document the date of consent in the subject's medical chart. Valid informed consent form is the most current version approved by the IRB. Each informed consent form should contain a subject authorization section that describes the uses and disclosures of a subject's personal information (including personal health information) that will take place in connection with the trial. If an informed consent / form does not include such a subject authorization, then the Investigator must obtain a separate subject authorization form from each subject.
- 9. Prepare and maintain adequate case histories of all persons entered into the trial, including eCRFs, hospital records, laboratory results, etc, and maintain these data for a minimum of 2 years following notification by the Sponsor that all investigations have been discontinued or that the regulatory authority has approved the marketing application. The Investigator should contact and receive written approval from the Sponsor before disposing of any such documents.
- 10. Allow possible inspection and copying by the regulatory authority of GCP-specified essential documents.
  - 11. Maintain current records of the receipt, administration, and disposition of Sponsor-supplied vaccines, and return all unused Sponsor-supplied vaccines to the Sponsor.

# APPENDIX B INVESTIGATOR CONSENT TO USE OF PERSONAL INFORMATION

Takeda will collect and retain personal information of Investigator, including his or her name, address, and other personally identifiable information. In addition, Investigator's personal information may be transferred to other parties located in countries throughout the world (eg, the United Kingdom, United States, and Japan), including the following:

- Takeda, its affiliates, and licensing partners.
- Business partners assisting Takeda, its affiliates, and licensing partners.
- Regulatory agencies and other health authorities.
- IRBs.

Investigator's personal information may be retained, processed, and transferred by Takeda and these other parties for research purposes including the following:

- Assessment of the suitability of Investigator for the trial and/or other clinical trials.
- Management, monitoring, inspection, and audit of the trial.
- Analysis, review, and verification of the trial results.
- Safety reporting and pharmacovigilance relating to the trial.
- Preparation and submission of regulatory filings, correspondence, and communications to regulatory agencies relating to the trial.
- Preparation and submission of regulatory filings, correspondence, and communications to regulatory agencies relating to other vaccines used in other clinical trials that may contain the same chemical compound present in the investigational vaccine.
- Inspections and investigations by regulatory authorities relating to the trial.
- Self-inspection and internal audit within Takeda, its affiliates, and licensing partners.
- Archiving and audit of trial records.
- Posting Investigator site contact information, trial details and results on publicly accessible clinical trial registries, databases, and websites.

Investigator's personal information may be transferred to other countries that do not have data protection laws that offer the same level of protection as data protection laws in Investigator's own country. Investigator acknowledges and consents to the use of his or her personal information by Takeda and other parties for the purposes described above.

- CONSENT FORM

  Conserved to each subject:

  Conserved to eac or placebo.
- 10. A description of the possible side effects following vaccine administration that the subject may receive.
- 11. A description of any reasonably foreseeable risks or discomforts to the subject and, when applicable, to an embryo, fetus, or nursing infant.
- 12. A statement that the vaccinations may involve risks to the subject (or to the embryo or fetus, if the subject is or may become pregnant) which are currently unforeseeable.
- 13. A description of any benefits to the subject or to others that reasonably may be expected from the research. When there is no intended clinical benefit to the subject, the subject should be made aware of this.
- 14. Disclosures of appropriate alternative procedures or courses of treatment, if any, that might be advantageous to the subject and their important potential risks and benefits.
- 15. A statement describing the extent to which confidentiality of records identifying the subject will be maintained, and a note of the possibility that regulatory agencies, auditor(s), IRB, and the monitor may inspect the records. By signing a written informed consent form, the subject is authorizing such access.
- 16. For research involving more than minimal risk, an explanation as to whether any compensation and an explanation as to whether any medical treatments are available if injury occurs and, if so, what they consist of or where further information may be obtained.
- 17. The anticipated prorated payment(s), if any, to the subject for participating in the trial.
- 18. The anticipated expenses, if any, to the subject for participating in the trial.

- 19. An explanation of whom to contact for answers to pertinent questions about the research (Investigator), subject's rights, and IRB and whom to contact in the event of a research-related injury to the subject.
- 20. A statement that participation is voluntary, that refusal to participate will involve no penalty or loss of benefits to which the subject otherwise is entitled, and that the subject may discontinue participation of their child at any time without penalty or loss of benefits to which the subject is otherwise entitled.
- 21. The consequences of a subject's decision to withdraw from the research and procedures for orderly termination of participation by the subject.
- 22. A statement that the subject will be informed in a timely manner if information becomes available that may be relevant to the subject's willingness to continue participation in the trial.
- 23. A statement that results of pharmacogenomic analysis will not be disclosed to an individual, unless prevailing laws require the Sponsor to do so.
- 24. The foreseeable circumstances or reasons under which the subject's participation in the trial may be terminated.
- 25. A written subject authorization (either contained within the informed consent form or provided as a separate document) describing to the subject the contemplated and permissible uses and disclosures of the subject's personal information (including personal health information) for purposes of conducting the trial. The subject authorization must contain the following statements regarding the uses and disclosures of the subject's personal information:
  - a) that personal information (including personal health information) may be processed by or transferred to other parties in other countries for clinical research and safety reporting purposes, including, without limitation, to the following: (1) Takeda, its affiliates, and licensing partners; (2) business partners assisting Takeda, its affiliates, and licensing partners; (3) regulatory agencies and other health authorities; and (4) IRBs;
  - b) it is possible that personal information (including personal health information) may be processed and transferred to countries that do not have data protection laws that offer subjects the same level of protection as the data protection laws within this country; however, Takeda will make every effort to keep your personal information confidential, and your name will not be disclosed outside the clinic unless required by law;
  - c) that personal information (including personal health information) may be added to Takeda's research databases for purposes of developing a better understanding of the safety and effectiveness of the investigational vaccine(s), studying other therapies for patients, developing a better understanding of disease, and improving the efficiency of future clinical trials;
  - d) that subjects agree not to restrict the use and disclosure of their personal information (including personal health information) upon withdrawal from the trial to the extent that

the restricted use or disclosure of such information may impact the scientific integrity of the research; and

- e) that the subject's identity will remain confidential in the event that trial results are published.
- 26. Female subjects of childbearing potential (eg, non-sterilized, premenopausal female subjects) who are sexually active must use adequate contraception (as defined in the informed consent form) from at least 2 months prior to Day 1 (M0) up to 6 weeks post second dose at Day 90 (M3). Pregnancy tests will be performed prior to vaccination at Day 1 (M0) and Day 90 (M3). Additional pregnancy tests may be performed during the trial if deemed necessary by the Investigator. Females of childbearing potential who are sexually active will be reminded during trial visits to adhere to acceptable contraceptive methods (see Section 7.2) up to 6 weeks post second dose. If a subject is found to be pregnant during the trial, no further vaccine doses will be administered.

e ... al will be ... and sulfante only and sulfa A statement that clinical trial information from this trial will be publicly disclosed in a publicly

## APPENDIX D SEROLOGY PLAN

#### Table 16.a Serology Plan

| Timing | Blood volume | Assessments |
|---|---|---|
| Day 1 (M0), Day 120 (M4), and Day 270 (M9) | 5 mL | Dengue neutralizing antibodies (by MNT <sub>50</sub> ) |

M=month, MNT50=microneutralization test

as immunoge a sample at Day and a thought to the address of the and a thought and a thought a th Note: Blood samples for immunogenicity testing will only be collected from subjects included in the immunogenicity subset. Blood sampling at Day 1 (M0) should be taken prior to administration of the first trial dose. The blood sample at Day 120 (M4) should be

Signature Page for DEN-304 Protocol Amendment 2, Version 4.0, 29 October 2018 Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Demonstr

| | Approval | | PPD | | 16 Letille |
|---|---|---|---|---|---|
| | Approval | | PPD | | 30, |
| | Approval | | PPD | 7 | |
| | Approval | | PPD | | |
| Property | of Takedai. For | Document Numb | er: TAK-003-0116 | 0 v4.0 | |